## Cover page

## Official title:

Sustainable-psycho-nutritional intervention program and its effects on water and carbon footprint, metabolic biomarkers, and gut microbiota in Mexican population: study protocol of a m-Health randomized clinical trial

### **Brief Title:**

Sustainable-psycho-nutritional intervention program and its effects on health outcomes and the environment

Date of the document: March 27, 2022

NCT: not yet available

Ethics committee number: CUCBA/CEIC/CE/002/2022

Mariana Lares-Michel<sup>1,2\*</sup>, Fatima Ezzahra Housni<sup>1•</sup>, Zyanya Reyes-Castillo<sup>1</sup>, Jesús Francisco Rodríguez

Huertas<sup>2</sup>, Virginia Gabriela Aguilera Cervantes<sup>1</sup>, Rosa María Michel Nava<sup>3</sup>

1. Instituto de Investigaciones en Comportamiento Alimentario y Nutrición (IICAN), University Center of the

South, University of Guadalajara. Address: Av. Enrique Arreola Silva 883, Col. Centro. Zip Code: 49000, Cd.

Guzmán, Jalisco, México.

2. Institute of Nutrition and Food Technology "José Mataix Verdú", Biomedical Research Center, University

of Granada, Avenida del Conocimiento S/N. Parque Tecnológico de la Salud. Armilla,18071 Granada, Spain

3. Tecnológico Nacional de México, Campus Ciudad Guzmán. Address: Avenida Tecnológico 100, Col. Centro.

Zip Code: 49000. Ciudad Guzmán, México.

\*This study protocol is the Ph.D. thesis of the student Mariana Lares-Michel, who is currently registered as Ph.D.

student at the University of Guadalajara and the University of Granada under a double Ph.D. title program. Contact

e-mail: marianalares@correo.ugr.es, mariana.lmichel@alumnos.udg.mx

•Responsible researcher on ClinicalTrials.gov: fatima.housni@cusur.udg.mx

Note: This study protocol will be submitted to a scientific journal as a study protocol.

2

#### Abstract

Mexico is going through a major environmental and nutritional crisis, which is related to unsustainable dietary behaviors. Sustainable diets could solve both problems together. However, in Mexico and the world, an intervention program oriented to promoting sustainable diets has not been designed. This study protocol aims to design a 3-stages, 15 weeks, sustainable-psycho-nutritional digital intervention program whose objective is to promote the adherence of the Mexican population to a sustainable diet and to evaluate its effects on dietary water and carbon footprints, metabolic biomarkers, and gut microbiota of this population. The behavior change wheel model and the guide for digital interventions design will be followed. In stage 1, the program will be designed using the sustainable diets model, and the behavior change wheel model. A sustainable food guide, sustainable recipes, and food plans as well as a mobile application will be developed. In stage 2, the intervention will be carried out for 7 weeks, and a follow-up period of 7 weeks, in a sample of Mexican young adults (18 to 35 years) randomly divided into an experimental group (n=50) and a control group (n=50). The nutritional care process model will be used. Anthropometric, biochemical, clinical, dietary, environmental, socioeconomic level and cultural aspects, nutritional-sustainable knowledge, behavioral aspects, and physical activity will be considered. Thirteen behavioral objectives will be included using successive approaches in online workshops twice a week. The population will be monitored using the mobile application that will include behavioral change techniques. In stage 3, the effects of the intervention will be assessed on the dietary water and carbon footprint, lipid profile, serum glucose, and gut microbiota composition of the evaluated population. We expected to find improvements in health outcomes and a decrease in the dietary water and carbon footprints. With this study, the first theoreticalmethodological approach to the sustainable-psycho-nutrition approach will be generated.

**Keywords:** Sustainable Diets, Behavior Change, Gut Microbiota, Environmental Impact of Diets, Nutritional and Environmental Education, Mexican Population, Water Footprint, Carbon Footprint, Eating Behavior, m-Health.

#### 1. Introduction

The change from the traditional Mexican diet to a Western diet, generated by the nutritional transition, has not only generated prevalence's of more than 75% of metabolic alterations (obesity, type 2 diabetes, cardiovascular diseases, dyslipidemia) (1–3) and in the gut microbiota of the Mexican population (4), but it has also generated the water and carbon footprint of their diet to be the highest in the world with more than 8,000 Liters per person per day (L p<sup>-1</sup>d<sup>-1</sup>) (5) and 6.01 Kg CO<sup>2</sup>eq p<sup>-1</sup>d<sup>-1</sup> (6), respectively. This is linked to the aggravation of climate change, with increases of more than 1.0 °C in the average atmospheric temperatures (7) and the current water crisis that Mexico is going through, which affects 85% of the territory and has been referred to as the worst water drought in history, affecting the water supply of millions of Mexicans (1,8).

One of the proposals for the joint solution of these problems has been the adoption of sustainable and territorial diets, which in Mexico could be carried out through the recovery of its traditional diet, both pre-Hispanic and colonized, which, prepared with low-fat culinary techniques and low content of animal products, can be considered as an appropriate option from a nutritional, cultural, economic and environmental perspective, dimensions that must be present for a diet to be considered as sustainable (1,9–12).

However, to achieve the adoption of a particular diet, it is necessary to modify the eating behavior of the population (13–15). To modify both dietary and unsustainable behaviors in a population, there are multiple strategies, among which intervention programs have stood out (14,16,17). However, to date and both nationally and internationally, no intervention program whose objective is to promote both adequate nutrition to improve health and reduce the environmental impact of dietary behaviors, has been reported. This respecting cultural, social, economic, and psychological aspects of the population.

Based on the above, this study protocol aims to design a three-stage 15 weeks intervention program, based on the guide to designing interventions of the behavior change wheel model (14), which includes both nutritional and sustainability elements, in the sense of considering unsustainable dietary behaviors of the Mexican population, in addition to taking into account their social, cultural and economic aspects. In addition to these axes, the basis of behavioral modification intervention programs is psychology. Therefore, it is proposed to design a sustainable-psycho-nutritional intervention program, whose objective is to promote the adherence of the population to sustainable diets. But, in addition, it is proposed to evaluate its effects on environmental indicators, metabolic biomarkers, and gut microbiota, as well as clinical aspects and body composition in a Mexican population sample. Because of the effectiveness of technologies use in nutritional (18,19) and environmental (20,21) interventions,

the intervention program will be a digital one, for which a mobile application is being designed to evaluate and monitor the intervened population. Therefore, this will be a m-Health intervention program.

We hypothesized that a sustainable-psycho-nutritional intervention digital program can modify the eating behavior of a Mexican population group and guide it towards a sustainable diet, generating decreases in glucose levels, total cholesterol (TC), LDL cholesterol (LDL-C), and triglycerides (TG), and increases in HDL cholesterol (HDL-C) levels. Likewise, we hypothesized that this type of program can modify the composition of the gut microbiota of the population, promoting the proliferation of bacteria related to metabolic health; reduce the water and carbon footprint of the sample's diets; maintain adequate body fat levels in the population with an adequate body fat percentage or reduce them in the overweight or obese population; maintain blood pressure levels in the healthy population and lower them in the population with high blood pressure, and reduce the presence of acanthosis nigricans.

#### 2. Methods

It is proposed to carry out a quasi-experimental longitudinal study of three stages that will be related to each other.

### 2.1 Stage 1: Design of the program

A sustainable-psycho-nutritional intervention program will be designed based on the characteristics of a sustainable diet for the national context of Mexico, adaptable to any regional context. It will include a mobile application that is being designed for this project, which will include a sustainable food guide, sustainable-psycho-nutritional workshops, sustainable recipes and food plans, and behavioral change techniques. The program will be designed based on the sustainable diets model (12) and concept (9), the behavior change wheel model (14), the guideline for the development and evaluation of digital behavioral interventions in health care (19), and on the guide to designing interventions of the behavior change wheel, which incorporate 3 stages and 8 development steps (22).

#### 2.1.1 Mobile application design

A mobile application (app) will be developed in collaboration with software and mobile applications developers and will be based on the user-centered methodology (23), and on the guide for the design of digital interventions by West and Michie (24). It will contain the following behavioral modification techniques: education

through workshops videos (13); persuasion by sending messages of risks and benefits (25), encouragement and coercion using token economy (13), nudges by messaging (26), self-monitoring by graphical progress viewing (27,28), successive approaches by behavioral objectives addressing (13), and guides (14), through a sustainable food guide that will be designed by means of linear programming optimization (29,30) using MATLAB®, and graphic design programs such as Adobe Illustrator® and BioRender®. This guide will be designed based on the recommendations of the FAO for the development of dietary guidelines (31) and on the Mexican Food Equivalent System (32). For the token economy system, cut-off points will be established to be charged to the app (Supplementary Material 1). Additionally, educational workshops and meal plans will be designed, following the model of sustainable diets of Johnston et al. (12), and using the Nutriecology® Nutritional-Ecological software and the Nutrimind® Software for diet calculation. Likewise, the guidelines for the prescription of meal plans, menu design, and recipes for the Mexican population will be followed (33). Prior to the launch of the mobile application, its feasibility, acceptability, quality, and usability will be assessed. Also, it will be evaluated following the APEASE criteria, which include evaluating the 1) Affordability, 2) Practicability, 3) Effectiveness, and Costeffectiveness, 4) Acceptability, 5) Side-effects/safety, and 6) Equity.

### 2.1.2 Behavior change intervention design process

The process of design of the intervention is shown in Table 1. The process of understanding the behavior, including the problem definition (1–3,5,6), the selected target behaviors, and what needs to be modified from them (12,13,27,34–36) are described. Also, the selected intervention functions (37), as well as the selected policy categories from the behavior change wheel model, are presented.

Table 1. Design of the Sustainable-Psycho-Nutritional intervention program according to the behavior change wheel model and guide for interventions design

| Stage 1: Understand | the behavior |
|---|---|
| Stage 1: Understand to Step 1: Define the problem in behavioral terms | This step will be based on the available scientific evidence on the country's dietary and environmental situation, which reveals high prevalence's of overweight, obesity, and associated pathologies such as type 2 diabetes, dyslipidemia, and hypertension (1,2,6). Also, the highest values of dietary water and carbon footprints were found (5,6). These problems are mainly related to inadequate food consumption (which will be further detailed) and lack of physical activity (1). |
| Step 2: Select target behavior | The target behaviors will be lack of physical activity performance, inadequate consumption of Mexican foods and dishes, fruits and vegetables, whole grains, legumes, seeds and healthy fats, dairy products, eggs, fish and shellfish, chicken, red |
| Step 3: Specify the target behavior | meat (beef and pork, and, in some cases, goat and lamb) and processed, ultra-<br>processed foods and added and free sugars, as well as foods high in trans and saturated fats. |
| Step 4: Identify what needs to change | Targets behaviors will be established as a goal-setting strategy, which has been reported to be one of the most effective methods for modifying dietary behaviors (27). Also, they will be addressed as successive approximations toward a sustainable diet, another effective behavior change technique (13,33). Targets behaviors will be: |
| | <ol> <li>Increase physical activity.</li> <li>Increase the consumption of sustainable Mexican foods and dishes.</li> <li>Increase the consumption of fruits and vegetables.</li> <li>Increase the consumption of whole grains.</li> <li>Increase the consumption of legumes.</li> <li>Increase the intake of seeds and healthy fats.</li> <li>Reduce dairy consumption.</li> <li>Reduce the consumption of eggs.</li> <li>Reduce consumption of fish and shellfish.</li> <li>Reduce the consumption.</li> <li>Reduce the consumption of red (beef, pork, goat, and lamb) and processed meats.</li> <li>Reduce the consumption of ultra-processed foods.</li> <li>Reduce the intake of added and free sugars, as well as foods with a high content of trans and saturated fats.</li> </ol> |
| | All foods whose consumption will be promoted will be aligned with the sustainability characteristics for the Mexican context (12), on the recommendations of a healthy diet provided by the WHO (35), and on the model QC7G for food and nutrition education, that will specify which foods to select, in which quantities, when to consumed them and how to prepare them. In addition to when to perform physical activity, specifying type and duration (13). |
| Stage 2: Identify inte | |
| Step 5: Intervention functions | The intervention functions from the behavior change wheel model will be: education, persuasion, incentivization, and coercion. These will be verified in relation to the APEASE criterion Michie et al. (36). |

Table 1. Continuation: Design of the Sustainable-Psycho-Nutritional intervention program according to the behavior change wheel model and guide for interventions design

Stage 2: Identify intervention options

Step 6: Policy categories

The policy category of the behavior change wheel model will be the guidelines. Therefore, a nutritional-sustainable food guide will be designed, using linear programming optimization (29, 30), based on the FAO recommendations for the development of dietary guidelines (31), and covering the elements of the sustainable diets model (12) as follows: 1) Wellness and Health: ABCD; A: anthropometric and body composition data (body weight and height, BMI, percentage of body fat, visceral fat, muscle mass, waist, and hip circumference, as well as waist-hip ratio); B: biochemical data (serum glucose, lipid profile and gut microbiota); C: clinical data (signs of nutrient deficiencies, acanthosis nigricans, and blood pressure). 2) Biodiversity, environment, and climate: carbon footprint and gray water footprint. 3) Equity and fair trade: food prices and socioeconomic level of the population. 4) "Ecofriendly", local, and seasonal foods: green and blue water footprint, locally produced and seasonal foods. 5) Cultural heritage and skills: Traditional Mexican diet, Mexican Diet Quality Index Adapted (IACDMx), and nutritional education based on a traditional diet. 6) Food needs, nutrients, food security, and access: personalized food plan according to individual requirements, preferences, and contexts. Figure 1 shows an adaptation of the model of sustainable diets of Johnston et al. (12) for this protocol characteristics.

Subsequently, this nutritional-sustainable food guide will be accompanied by a system of equivalent foods (32) that, in addition to incorporating the food's nutrients, will integrate their environmental impact. The calculation of the environmental impact will be made based on the calculation of the total, green, blue, and gray water footprint, using the Water Footprint Assessment method for Mexico (5). Likewise, the greenhouse gas emissions of foods will be calculated, using the Life Cycle Assessment method for food production and processing through pre-quantified databases (55,56,57). The prices and cultural characteristics of the main consumed foods in Mexico will be included (5,32). Prices will be obtained based on fieldwork in supermarkets, and a review of supermarket databases, while cultural aspects will be determined based on a literature review of the traditional Mexican diet (1,10).

Once sustainability dimensions are calculated, a sustainable recipe book will be developed, including examples of food plans with individualization options. These food plans will be made up of a distribution of equivalent food rations (32) and examples of menus that meet the nutritional and sustainability characteristics of the Mexican population, with adaptations options.

### Stage 3: Identify content and implementation options

Step 7: Behavior change techniques

Specific behavior change techniques will be used covering the selected intervention functions as follows:

- Education: successive approximations in the workshops addressing the target objectives.
- Persuasion: Nudges, risk, and benefits communication.
- Incentivization, coercion, and monitoring: messaging, remainders, and token economy through food registers by writing and photos on the mobile application.
- Social support: forum in the mobile app where participants can share pictures
  of their foods and their physical activity performance. Also, will be able to like
  the photos of other participants and comment on the photos. Also, a chat for the
  resolution of doubts between user and administrator will be included in the
  mobile application.

Step 8: Mode of delivery

The mode of delivery will be digital since a mobile application is being designed and the workshops will be delivered by digital platforms in videos.



Figure 1. Sustainable-Psycho-Nutritional approach for the intervention design, based on the sustainable diets model (12), The behavior change wheel model (14), and the COM-B model (14). Own elaboration.

#### 2.2 Stage 2: Application of the sustainable-psycho-nutritional intervention program

#### 2.2.1 Participants

Once the intervention program has been designed, it will be applied to a sample of Mexican young adults from the south of Jalisco, randomly divided into two groups: an experimental group (n=50) and a control group (n=50). This is based on recommendations for group designs in behavior modification programs (38). The sample size is according to the minimum suggested for nutritional interventions (39,40), and taking into account the possible desertion of the participants during the intervention, which can amount to more than 50% of the initial sample (41). We will include a population between 18 and 35 years old, with Body Mass Index (BMI) values from 18.5 to 40, with or without risk factors for the development of chronic diseases, but without diagnosis with previous pharmacological treatment. The inclusion, exclusion, and elimination criteria are detailed in Supplementary Material 2 in Table SM2.1. Also, for being included in the study cut-off points to identify inadequate consumption and physical activity were established (Table SM2.2). The population will be invited to participate through social networks and posters at strategic points, such as Universities, gyms, and the downtown city. Young adults were selected as the population for this study since they are already considered adults who make autonomous food decisions, but at the same time, their young age makes them susceptible to behavioral modification. In addition, they represent parents or future parents, as well as the active population of Mexico, so providing nutritional-sustainable education to these people could generate long-term benefits for their health and that of their families (21,42,43).

#### 2.2.2 Procedure

Participants will be evaluated following the nutritional care process model (44). The first evaluation will be performed at the beginning of the intervention at baseline, and according to individual requirements, the behavioral objectives will be individually adapted and will be addressed for 7 weeks, considering 2 objectives per week, thus providing 2 weekly educational workshops. Also, personalized food plans will be prescribed, according to the linear programming optimization (29,30) performed at MATLAB®.

After 7 weeks of educational and nutritional intervention, at week 8, the experimental population will be divided into two sub-groups, where one group will stop being intervened completely (n = 25), and another will continue to receive messages through the mobile application (n = 25) for 8 weeks. Finally, at week 15, a final evaluation will be carried out. The study design is shown in Figure 2. Participants will be evaluated in the regard of Anthropometric, Biochemical, Clinical, Dietetics, Environmental, Socioeconomic level and cultural aspects,

Nutritional-sustainable knowledge, Behavioral aspects, and Physical activity (ABCD-ESNBP). These aspects will be evaluated according to the nutritional care process model, thus identifying the problem of the population, establishing the etiology, and stating the signs and symptoms (44).

#### 2.2.3 Sustainable-psycho-nutritional indicators

The ABCD-ESNBP indicators will be included in a complete clinical history that will be uploaded to the mobile application (Supplementary Material 3) and will be evaluated as follows: A) Anthropometric: height with a Smartmet® stadiometer, weight, and body composition (percentage of body fat, muscle mass, visceral fat) with an Omron® bioimpedance scale (HBF-511T-E/HBF-511B-E), BMI = weight/height², waist and hip circumference using a Lufkin® metal tape measure. The assessment will be performed following the validated techniques of Suverza and Haua (45).

B) Biochemical: glucose and lipid profiles (TC, LDL-C, HDL-C, and TG) will be determined through blood samples that will be taken from the antecubital vein of each participant, following the protocol from the Mexican Health Secretary (46,47). Samples will be taken by specialists, after an overnight fast of 8 to 12 hours and will be centrifuged at 3500 rpm for 15 min to separate the serum. Samples will be aliquoted and stored at -20°C until the day of testing. Tourniquets, alcohol swabs, 10 mL syringes, and blood collection tubes will be required. Gut microbiota will also be analyzed, for which fecal samples will be collected in a sterile stool container using a sterile kit including gloves and a spatula that will be delivered to the participants. Once collected, the samples will be divided into aliquots and will be stored at -80 °C, following a method used for the Mexican population (4,48).

C) Clinical: a clinical history will be carried out, covering pathologies suffering, pathological family history, medicaments, and supplement use (Supplementary Material 3). Clinical signs of insulin resistance (acanthosis nigricans) will be evaluated by physical exploration, searching for hyperpigmentation and thickening of the skin with velvety, in visible flex areas (axilla, anterior ulnar area, and posterior and lateral region of the neck) (49). Signs of nutrient deficiencies or excess will also be evaluated in relation to hair, nails, mouth, tongue, edema, and mucous membranes appearance (45). Likewise, blood pressure will be evaluated with a Medstar® sphygmomanometer and following the Mexican normativity (50).



Note. ABCD-ESNBP: Anthropometric, Biochemical, Clinical, Dietetics, Environmental, Socioeconomic level and cultural aspects, Nutritional-sustainable knowledge, Behavioral aspects, and Physical activity.

Figure 2. Study design for stage 2. Own elaboration.

- D) Dietetics: caloric-nutritional intake will be assessed through 24-hour recalls and dietary records (51), and by a validated adapted Food Frequency Questionnaire (CFCA) (5,52). Diet quality will also be analyzed by an adapted version of the Mexican Diet Quality Index (ICDMx) (53). Participants will also be asked about food preparation, food shopping places, food allergies and intolerances, food preferences, and about following specific diets at the moment of the evaluation.
- E) Environmental: dietary water footprint will be calculated using the Water Footprint Assessment method (54) in its version for Mexico's context (5). The water footprint of each food and food ingredients are going to be calculated. Also, water involved in cooking and food washing is going to be evaluated. Dietary carbon footprint is also going to be calculated using the Life Cycle Assessment method (7,55,56). Food system boundaries are going to be the impact of food production and processing on greenhouse gas emissions, as carried out by Fresán et al. (57). Corrections factors from converting cooked to uncooked food and peeled to unpeeled food are going to be applied. Both calculations are going to be performed in the Nutriecology® Software.
- S) Socioeconomic level and cultural aspects: educational level, occupational level, and economic income are going to be evaluated according to classifications used for Mexico, which are detailed in Supplementary Material 3 (58). For this aspect, food prices are going to be investigated in fieldwork and in supermarket databases, in order to promote the consumption of accessible foods. Also, food culture related to celebrations and traditions is going to be investigated.
- N) Nutritional-sustainable knowledge: it will be evaluated through a designed questionnaire (Supplementary Material 4), based on the psychological capacity presented in the COM-B model. It will include a series of questions for the evaluation of nutritional-sustainable knowledge, which will be related to the established behavioral objectives and will be based on manuals for the design of nutritional knowledge questionnaires and on questions on sustainable food consumption (59–62).
- B) Behavioral aspects: all dimensions of the COM-B model will be assessed in a designed questionnaire based on Brain et al. (63) (Supplementary Material 4). The questions will be related to physical and psychological ability, automatic and reflexive motivation, and physical and social opportunity (14). Questions were adapted according to the context of sustainable diets (12): (1) Capacity: knowledge of sustainable nutrition, preparation skills food and preparation capacity; (2) Opportunity: time to eat and prepare food, access to food, and food storage; (3) Motivation: the desire to change eating habits, emotions involved in food consumption and habits that participants are willing to change.

P) Physical activity: the IPAQ questionnaire will be used, which is included in the clinical history shown in Supplementary Material 3. Besides the questionnaire, specific questions about physical activity type, frequency, intensity, and duration are going to be asked.

#### 2.3 Stage 3: Effects of the sustainable-psycho-nutritional intervention program

As the last stage of this protocol, the corresponding laboratory analyses, and statistical tests will be carried out.

#### 2.3.1 Metabolic biomarkers analysis

For the analysis of metabolic biomarkers, colorimetric enzymatic methods will be used using the Spinreact® S. A/S A. U (Girona, Spain) laboratory kits, for fasting glucose determination (Cat. No. 1001190), TC (Cat. No. 41022), LDL-C (Cat. No. BSIS51-E), HDL-C (Cat. No. BSIS37-E) and TG (Cat. No. 1001313) (47). The reference points for glucose values and lipid profiles will be taken from the regulations in force in Mexico (64,65).

#### 2.3.2 Gut microbiota analysis

For the analysis of the gut microbiota, the real-time quantitative polymerase chain reaction (qPCR) method will be followed (4,48). First, DNA will be extracted from the collected stool samples, following the protocol for rapid purification of genomic DNA from stool samples. The Qiagen brand commercial kit (1066790ES, USA) will be used. This procedure integrates two stages: lysis and separation of impurities from stool samples, for which Inhibitex Buffer will be used and DNA purification will be carried out by means of centrifugation columns. Once the bacterial DNA samples are obtained, they will be stored and labeled in sterile plastic microtubes (Eppendorf 1.6 mL) at a temperature of -80°C until further analysis.

Next, the purity of the DNA will be verified, and its concentration will be determined using a NanoDrop Lite spectrophotometer (Thermo Scientific, Waltham, MA, USA). 1  $\mu$ L of the DNA stock of each sample will be placed on the lens of the equipment and the sample will be read at a wavelength of 260 nm for DNA quantification and at 280 nm for protein quantification. The purity will be determined by calculating the index performed by the team, by dividing the reading at 260 nm by the reading at 280 nm and will be considered acceptable in a range of 1.5 to 2. The concentration of the purified coproDNA sample will be measured by their absorbance ratio of 260/280 nm using the same spectrophotometer. This analysis corresponds to the absorbance index of nucleic acids and provides the final concentration in  $ng/\mu$ L (4,48,66).

Once the previous analyzes have been completed, the identification of the gut microbiota will be carried out using the qPCR molecular technique, on the StepOne Applied BioSystems platform, using the SYBR Green reagent as DNA detection chemistry. This reagent is considered an agent that intercalates into the DNA double helix and fluoresces as the DNA copies are synthesized. Therefore, at a higher concentration of the DNA of interest (bacterial), the equipment will record a higher fluorescence signal. In this case, the analysis of interest will be carried out in the V3-V4 hypervariable region of the bacterial 16S rRNA gene. For this analysis, specific primers, which are detailed in Supplementary Material 5 will be used. The bacterial load and relative abundance of the main bacteria present in the intestine (Firmicutes and Bacteroidetes) (4,67,68) will be determined, as well as those related to particular types of diets, for example, Lactobacillus and Bifidobacterium that are related to healthy, vegetarian and Mediterranean diets (67,69,70), Faecalibacterium prausnitzii that is related to healthy diets and an anti-inflammatory effect (41,71–73), as well as Akkermansia muciniphila, which besides of being related to anti-inflammatory effects is associated to the consumption of the Mexican pre-Hispanic diet (41,70,72,74,75). The presence of Prevotella copri will also be identified, which is one of the bacteria most related to plant-based diets and is considered anti-inflammatory and glucose modulator (75,76). The presence of Bilophila wadsworthia will also be identified, as it is related to diets with a high content of foods of animal origin, mainly dairy and meat (71,77), as well as in westernized diets (67,78). Likewise, the presence of Clostridium coccoides will be analyzed, as it is related to obesity (48) and a high fat intake (79). Also, Streptococcus thermophilus will be included because it is related to dairy consumption (71,80). The exact procedure to follow regarding the qPCR run, as well as the specific conditions and temperatures of the analysis, are presented in the investigation of Rodríguez-Lara et al. (48), which will serve as the guide for this research project.

### 2.3.3 Evaluation of the adherence to the program

To measure the adherence of the intervened population to the program, an adapted questionnaire will be applied based on that of Gila-Díaz et al. (81), which will consist of the contrast of the recommendations provided with the performance of the behaviors to promote. For example, questions about the type and intensity of physical activity performed and the amount and frequency of consumption of each of the foods included in the behavioral objectives will be included. This questionnaire is shown in Supplementary Material 6.

#### 2.3.4 Statistical analyses

The distribution of the data will be analyzed with the Kolmogorov Smirnov test. Descriptive analysis will be performed, including means, standard deviations, and medians. Next, the effects of the program on the selected variables will be assessed by comparing them between evaluations and between groups with t-student tests for paired and unpaired data, respectively, if a normal distribution is found. For no normally distributed data, the Wilcoxon test (repetitive measures) and the U de Mann Whitney test (independent groups) will be used. For no categorical variables, the chi-squared test will be used. Correlation analyses will also be performed, considering Pearson correlation for normally distributed data and Spearman correlations for no normally distributed data. Likewise, simple, and multiple linear regression models will be carried out, as well as binary logistic regression analysis, to identify relationships and risks between variables. Statistical analysis will be performed at STATA V12® program.

#### 2.4 Ethical and biosafety considerations

This project has been already evaluated and approved by the Ethics Committee of the Center for Studies and Research in Behavior, of the University Center for Biological and Agricultural Sciences (CUCBA) from the University of Guadalajara with the number CUCBA/CEIC/CE/002/2022 and by the Technical Research Committee of the University Center of the South (CUSUR), with the number 2021D001. This protocol will also be registered on Clinical Trials.gov. When performing the intervention, the Declaration of Helsinki (82) and biosafety protocols of the Secretary of Health of Mexico (83) will be followed all the time. All participants will sign an informed consent (Supplementary Material 7) and their identities will be protected by the Federal Law on Protection of Personal Data Held by Private Parties (84).

Both due to regulations in research with human beings, and due to the situation of the COVID-19 pandemic, a strict biosafety protocol will be followed, where mouth covers will be always worn, both by the evaluating staff and by the participants. Likewise, the sample collection personnel will wear protective glasses and sterile gloves and constant disinfection of the work area will be carried out. In addition, hazardous biological waste will be disposed of in a special trash can in accordance with the provisions of the Ministry of Health (85).

#### 3. Discussion

By developing this program, we would be generating the first bases for the Mexican population (and future populations) to achieve a healthy and sustainable diet that can have positive effects on health outcomes and decrease the environmental impact of food consumption; thus addressing two of the main problems afflicting the

world population. Also, we are proposing a new concept: The Sustainable-Psycho-Nutrition, which is proposed as an approach based on behavioral science that integrates the psychological, social, cultural, economic, nutritional, and environmental aspects of eating behavior, whose objective is to generate the necessary bases to carry out behavioral change interventions, to guide the eating behavior of the population, towards sustainable eating behaviors. Within this term, we also launch the nutritional-ecological education, whose objective is to get people to acquire and performed the appropriate behavioral repertoire to determine what, how much, when, and how to eat, in relation to when, how much, and how energy is spent to maintain or recover their physical well-being, considering at all times the environmental impact of their behaviors and selecting the most sustainable foods, regarding the environment, culture, economy, preferences, food security, health, nutrition, among other factors (13).

Besides those aspects, the mobile application that we are currently developing is going to be a tool that will facilitate the promotion of sustainable diets first at the national level in Mexico, and forward, worldwide. Also, we will generate the first sustainable food guide for Mexico's context that will consider not only sustainability aspects but psychological and behavioral aspects. Moreover, the workshops, recipes, and food plans that we are creating are going to serve as tools for the health and environmental sector of the country to promote the consumption of sustainable diets. Finally, the link between gut microbiota and sustainable diets is a new aspect that this study will be characterized for the first time, specifically for the Mexican population. Finally, this project intends to bring attention to the importance of considering behavioral interventions and techniques for promoting sustainable diets.

#### References

- Lares-Michel M, Housni FE, Aguilera Cervantes VG, Reyes-Castillo Z, Michel Nava RM, Llanes Cañedo C, López Larios M de J. The water footprint and nutritional implications of diet change in Mexico: a principal component analysis. Eur J Nutr 2022;
- 2. Encuesta Nacional de Salud y Nutrición (ENSANUT). Encuesta Nacional de Salud y Nutrición [Internet]. 2018 [cited 2021 Jan 27]. Available from: https://ensanut.insp.mx/encuestas/ensanut2018/informes.php
- 3. Lares-Michel M, Housni FE, Aguilera Cervantes VG, Carrillo P, Michel Nava RM, Cañedo CL. Eat well to fight obesity... and save water: The water footprint of different diets and caloric intake and its relationship with adiposity. Front Nutr [Internet] Frontiers; 2021 [cited 2021 Jun 21];8. Available from: https://www.frontiersin.org/articles/10.3389/fnut.2021.694775/full
- Chávez-Carbajal A, Nirmalkar K, Pérez-Lizaur A, Hernández-Quiroz F, Ramírez-Del-Alto S, García-Mena J, Hernández-Guerrero C. Gut Microbiota and Predicted Metabolic Pathways in a Sample of Mexican Women Affected by Obesity and Obesity Plus Metabolic Syndrome. Int J Mol Sci 2019;20:E438.

- 5. Lares-Michel M, Housni FE, Aguilera Cervantes VG. A quantitative estimation of the water footprint of the Mexican diet, corrected for washing and cooking water. Food Sec 2021;13:849–74.
- 6. Magkos F, Tetens I, Bügel SG, Felby C, Schacht SR, Hill JO, Ravussin E, Astrup A. The Environmental *Foodprint* of Obesity. Obesity [Internet] 2020 [cited 2022 May 10];28:73–9. Available from: https://onlinelibrary.wiley.com/doi/10.1002/oby.22657
- 7. Willett W, Rockström J, Loken B, Springmann M, Lang T, Vermeulen S, Garnett T, Tilman D, DeClerck F, Wood A, et al. Food in the Anthropocene: the EAT–Lancet Commission on healthy diets from sustainable food systems. The Lancet [Internet] Elsevier; 2019 [cited 2021 Jan 27];393:447–92. Available from: https://www.thelancet.com/journals/lancet/article/PIIS0140-6736(18)31788-4/abstract
- 8. Sequía generalizada en México | Ciencia de la NASA [Internet]. [cited 2022 Jan 21]. Available from: https://ciencia.nasa.gov/sequia-generalizada-en-mexico?fbclid=IwAR03EyrjUZNenrcgXIsLaF4SKXfPbS4A5RE9Zs82DrWdy\_ADZ0itDt5pbfc
- 9. Food and Agriculture Organization of the United Nations, World Health Organization. Sustainable healthy diets: guiding principles. [Internet]. 2019 [cited 2021 May 14]. Available from: http://www.fao.org/3/ca6640en/ca6640en.pdf
- Valerino-Perea S, Lara-Castor L, Armstrong MEG, Papadaki A. Definition of the Traditional Mexican Diet and Its Role in Health: A Systematic Review. Nutrients [Internet] Multidisciplinary Digital Publishing Institute; 2019 [cited 2021 Jan 27];11:2803. Available from: https://www.mdpi.com/2072-6643/11/11/2803
- 11. Almaguer González J, García Ramírez H, Padilla Mirazo M, González Ferral M. Fortalecimiento de la salud con comida, ejercicio y buen humor: La dieta de la milpa. Modelo de alimentación mesoamericana saludable y culturalmente pertinente. Secretaría de Salud. [Internet]. Google Docs. 2019 [cited 2021 Jan 27]. Available from: https://drive.google.com/file/d/1n05pSVGY09FlzW91Rt8IZk\_6J-KIPRJT/view?usp=sharing&usp=embed facebook
- 12. Johnston JL, Fanzo JC, Cogill B. Understanding sustainable diets: a descriptive analysis of the determinants and processes that influence diets and their impact on health, food security, and environmental sustainability. Adv Nutr 2014;5:418–29.
- 13. López-Espinoza A, Martínez Moreno AG. La Educación en Alimentación y Nutrición. 2016.
- 14. Michie S, van Stralen MM, West R. The behaviour change wheel: A new method for characterising and designing behaviour change interventions. Implementation Science [Internet] 2011 [cited 2022 May 10];6:42. Available from: https://doi.org/10.1186/1748-5908-6-42
- 15. López-Espinoza A, Magaña González C. Hábitos Alimentarios: Psicobiología y socioantropología de la alimentación. 2014.
- 16. Vijayapushpam T, Antony GM, Rao GMS, Rao DR. Nutrition and health education intervention for student volunteers: topic-wise assessment of impact using a non-parametric test. Public Health Nutr 2010;13:131–6.
- North American Association for Environmental Education [NAAEE] / Secretaría de Medio Ambiente y Recursos Naturales [SEMARNAT] [NAAEE/SEMARNAT]. Guía para elaborar programas de educación ambiental no formal. [Internet]. 2009 [cited 2022 Jun 10]. Available from: https://biblioteca.semarnat.gob.mx/janium/Documentos/Ciga/libros2009/CG009094.pdf
- 18. Gabrielli S, Dianti M, Maimone R, Betta M, Filippi L, Ghezzi M, Forti S. Design of a Mobile App for Nutrition Education (TreC-LifeStyle) and Formative Evaluation With Families of Overweight Children. JMIR Mhealth Uhealth 2017;5:e48.
- 19. West R, Michie S. A Guide to Development and Evaluation of Digital Behaviour Change Interventions in Healthcare. London; 2016.

- Hedin B, Katzeff C, Eriksson E, Pargman D. A Systematic Review of Digital Behaviour Change Interventions for More Sustainable Food Consumption. Sustainability [Internet] Multidisciplinary Digital Publishing Institute; 2019 [cited 2022 Jun 10];11:2638. Available from: https://www.mdpi.com/2071-1050/11/9/2638
- 21. Pieniak Z, Żakowska-Biemans S, Kostyra E, Raats M. Sustainable healthy eating behaviour of young adults: towards a novel methodological approach. BMC Public Health 2016;16:577.
- 22. The Behaviour Change Wheel Book A Guide To Designing Interventions [Internet]. [cited 2022 May 10]. Available from: http://www.behaviourchangewheel.com/
- 23. Mor E, Garreta M, Galofré M. Diseño Centrado en el Usuario en Entornos Virtuales de Aprendizaje, de la Usabilidad a la Experiencia del Estudiante. :10.
- 24. A Guide to Development and Evaluation of Digital Behaviour Change Interventions in Healthcare Buy now at Silverback Publishing [Internet]. [cited 2022 May 10]. Available from: https://silverbackpublishing.org/products/cbc-monograph-1
- Spiegelhalter D. Risk and Uncertainty Communication. Annual Review of Statistics and Its Application [Internet] 2017 [cited 2022 Jun 6];4:31–60. Available from: https://doi.org/10.1146/annurev-statistics-010814-020148
- 26. Friis R, Skov LR, Olsen A, Appleton KM, Saulais L, Dinnella C, Hartwell H, Depezay L, Monteleone E, Giboreau A, et al. Comparison of three nudge interventions (priming, default option, and perceived variety) to promote vegetable consumption in a self-service buffet setting. PLoS One 2017;12:e0176028.
- 27. Rr R, Lj M, K H, Lt W. The Use of Behavior Change Theories in Dietetics Practice in Primary Health Care: A Systematic Review of Randomized Controlled Trials. Journal of the Academy of Nutrition and Dietetics [Internet] J Acad Nutr Diet; 2020 [cited 2022 Jun 7];120. Available from: https://pubmed.ncbi.nlm.nih.gov/32444328/
- 28. Spahn JM, Reeves RS, Keim KS, Laquatra I, Kellogg M, Jortberg B, Clark NA. State of the evidence regarding behavior change theories and strategies in nutrition counseling to facilitate health and food behavior change. J Am Diet Assoc 2010;110:879–91.
- 29. Gazan R, Brouzes CMC, Vieux F, Maillot M, Lluch A, Darmon N. Mathematical Optimization to Explore Tomorrow's Sustainable Diets: A Narrative Review. Adv Nutr 2018;9:602–16.
- 30. Maillot M, Vieux F, Amiot MJ, Darmon N. Individual diet modeling translates nutrient recommendations into realistic and individual-specific food choices. Am J Clin Nutr 2010;91:421–30.
- 31. Guías alimentarias y sostenibilidad [Internet]. Food and Agriculture Organization of the United Nations. [cited 2022 Jun 10]. Available from: http://www.fao.org/nutrition/educacion-nutricional/food-dietary-guidelines/background/sustainable-dietary-guidelines/es/
- 32. Pérez-Lizaur AB, Berenice Palacios González, Ana Laura Castro Becerra, Isabel Flores Galicia. Sistema Mexicano de Alimentos Equivalentes. Ogali; 2014.
- 33. Bertha P-L Ana Bertha. Desarrollo del Plan alimentario. Dietas normales y terapéuticas: los alimentos en la salud y la enfermedad. Sexta edición. 2014. p. 1–14.
- 34. Martínez Moreno AG. Control conductual y obesidad infantil. México obeso: actualidades y perspectivas. Editorial Universitaria. 2015. p. 238–49.
- 35. Martínez-Moreno AG. Modificación de la conducta alimentaria. Una asignatura para nutriólogos. La educación en alimentación y nutrición. [Internet] McGraw Hill. [cited 2022 Jun 10]. p. 253–66. Available from: https://www.researchgate.net/profile/Alma-Gabriela-Martinez-Moreno

- 36. World Health Organization [WHO]. Healthy diet. Fact Sheet N°394. [Internet]. 2015 [cited 2022 Jun 10]. Available from: https://www.who.int/publications/m/item/healthy-diet-factsheet394
- 37. Michie S, Atkins L, West R. The behaviour change wheel: a guide to designing interventions. 2014.
- 38. Gutierrez A. Modificacion de la conducta y sus aplicaciones Alan Kazdin pdf(cut). [cited 2022 Jun 8]; Available from: https://www.academia.edu/40179871/Modificacion\_de\_la\_conducta\_y\_sus\_aplicaciones\_Alan\_Kazdin\_p df\_cut\_
- 39. Duthie SJ, Duthie GG, Russell WR, Kyle JAM, Macdiarmid JI, Rungapamestry V, Stephen S, Megias-Baeza C, Kaniewska JJ, Shaw L, et al. Effect of increasing fruit and vegetable intake by dietary intervention on nutritional biomarkers and attitudes to dietary change: a randomised trial. Eur J Nutr 2018;57:1855–72.
- 40. Päivärinta E, Itkonen ST, Pellinen T, Lehtovirta M, Erkkola M, Pajari A-M. Replacing Animal-Based Proteins with Plant-Based Proteins Changes the Composition of a Whole Nordic Diet-A Randomised Clinical Trial in Healthy Finnish Adults. Nutrients 2020;12:E943.
- 41. Medina-Vera I, Sanchez-Tapia M, Noriega-López L, Granados-Portillo O, Guevara-Cruz M, Flores-López A, Avila-Nava A, Fernández ML, Tovar AR, Torres N. A dietary intervention with functional foods reduces metabolic endotoxaemia and attenuates biochemical abnormalities by modifying faecal microbiota in people with type 2 diabetes. Diabetes Metab 2019;45:122–31.
- 42. Petry N M. A comparison of young, middle-aged, and older adult treatment-seeking pathological gamblers PubMed. Gerontologist [Internet] [cited 2021 Jun 22];42:92–9. Available from: https://pubmed.ncbi.nlm.nih.gov/11815703/
- 43. Swinburn BA, Caterson I, Seidell JC, James WPT. Diet, nutrition and the prevention of excess weight gain and obesity. Public Health Nutr 2004;7:123–46.
- 44. Swan WI, Vivanti A, Hakel-Smith NA, Hotson B, Orrevall Y, Trostler N, Beck Howarter K, Papoutsakis C. Nutrition Care Process and Model Update: Toward Realizing People-Centered Care and Outcomes Management. J Acad Nutr Diet 2017;117:2003–14.
- 45. Suverza A, Haua K. El ABCD de la evaluación del estado de nutrición [Internet]. 1th ed. McGraw-Hill; 2010 [cited 2021 Jan 27]. Available from: https://issuu.com/jcmamanisalinas/docs/el abcd de la evaluaci n del estad
- 46. Peñalosa MAA. Norma Oficial Mexicana NOM-253-SSA1-2012, Para la disposición de sangre humana y sus componentes con fines terapéuticos. 2012;140.
- 47. Porchas-Quijada M, Reyes-Castillo Z, Muñoz-Valle JF, Durán-Barragán S, Aguilera-Cervantes V, López-Espinoza A, Vázquez-Del Mercado M, Navarro-Meza M, López-Uriarte P. IgG Anti-ghrelin Immune Complexes Are Increased in Rheumatoid Arthritis Patients Under Biologic Therapy and Are Related to Clinical and Metabolic Markers. Front Endocrinol (Lausanne) 2019;10:252.
- 48. Rodríguez-Lara A, Plaza-Díaz J, López-Uriarte P, Vázquez-Aguilar A, Reyes-Castillo Z, Álvarez-Mercado AI. Fiber Consumption Mediates Differences in Several Gut Microbes in a Subpopulation of Young Mexican Adults. Nutrients [Internet] Multidisciplinary Digital Publishing Institute; 2022 [cited 2022 Jun 7];14:1214. Available from: https://www.mdpi.com/2072-6643/14/6/1214
- Pinheiro AC, Rojas P, Carrasco F, Gómez P, Mayas N, Morales I. Acanthosis nigricans as an indicator of insulin resistance in Chilean adult population. Nutrición Hospitalaria [Internet] 2011 [cited 2022 Jun 8];26:940–4. Available from: http://scielo.isciii.es/scielo.php?script=sci\_abstract&pid=S0212-16112011000500003&lng=es&nrm=iso&tlng=en
- 50. NOM-030-SSA2-2009, Para la prevención, detección, diagnóstico, tratamiento y control de la hipertensión arterial sistémica. | Comisión Nacional de los Derechos Humanos México [Internet]. [cited

- 2022 Jun 7]. Available from: https://www.cndh.org.mx/documento/nom-030-ssa2-2009-para-la-prevencion-deteccion-diagnostico-tratamiento-y-control-de-la
- 51. Rosa M. Ortega CP-R Ana M López-Sobaler,-. Métodos de evaluación de la ingesta actual: registro o diario diétetico. REVISTA ESPAÑOLA DE NUTRICION COMUNITARIA [Internet] 2015 [cited 2022 Jun 7];34–41. Available from: https://doi.org/10.14642/RENC.2015.21.sup1.5048
- 52. Macedo-Ojeda G, Vizmanos-Lamotte B, Márquez-Sandoval YF, Rodríguez-Rocha NP, López-Uriarte PJ, Fernández-Ballart JD. Validation of a semi-quantitative food frequency questionnaire to assess food groups and nutrient intake. Nutr Hosp 2013;28:2212–20.
- 53. Macedo-Ojeda G, Márquez-Sandoval F, Fernández-Ballart J, Vizmanos B. The Reproducibility and Relative Validity of a Mexican Diet Quality Index (ICDMx) for the Assessment of the Habitual Diet of Adults. Nutrients 2016;8.
- 54. Hoekstra AY, Chapagain AK, Aldaya MM, Mekonnen MM. The Water Footprint Assessment Manual: Setting the Global Standard [Internet]. 1st ed. Routledge; 2012 [cited 2021 Jan 27]. Available from: https://www.taylorfrancis.com/books/9781849775526
- 55. Green RF, Joy EJM, Harris F, Agrawal S, Aleksandrowicz L, Hillier J, Macdiarmid JI, Milner J, Vetter SH, Smith P, et al. Greenhouse gas emissions and water footprints of typical dietary patterns in India. Sci Total Environ 2018;643:1411–8.
- 56. Ruiz Cerrillo S. Modelo de cálculo de la huella de carbono para el sistema Mexicano de alimentos equivalentes. JOURNAL OF NEGATIVE AND NO POSITIVE RESULTS [Internet] 2017 [cited 2022 Jun 10];226–32. Available from: https://doi.org/10.19230/jonnpr.1240
- 57. Fresán U, Martínez-Gonzalez M-A, Sabaté J, Bes-Rastrollo M. The Mediterranean diet, an environmentally friendly option: evidence from the Seguimiento Universidad de Navarra (SUN) cohort. Public Health Nutr 2018;21:1573–82.
- 58. Lares-Michel M, Housni FE, Cervantes VGA, Cañedo CL, Carmona M del CB, Toro HBD, Nava RMM. The Relationship between Consumption, Socioeconomic Level and Reasons of Tomato Intake in Mexico. Agricultural Sciences [Internet] Scientific Research Publishing; 2018 [cited 2021 Jan 27];9:720–6. Available from: https://m.scirp.org/papers/abstract/85913
- 59. The Kap Survey model Knowledge attitude and practices [Internet]. [cited 2022 Jun 8]. Available from: https://www.medecinsdumonde.org/en/actualites/publications/2012/02/20/kap-survey-model-knowledge-attitude-and-practices
- 60. World Health Organization, Partnership ST. Advocacy, communication and social mobilization for TB control: a guide to developing knowledge, attitude and practice surveys [Internet]. World Health Organization; 2008. Report No.: WHO/HTM/STB/2008.46. Available from: https://apps.who.int/iris/handle/10665/43790
- 61. Fautsch Y, Glasauer P, Nutrition Division. Guidelines for assessing nutrition-related knowledge, attitudes and practices [Internet]. Rome, Italy: FAO; 2014 [cited 2022 Jun 8]. 188 p. Available from: https://www.fao.org/publications/card/es/c/e1dfc1bb-0951-5221-a333-961243626fb6/
- 62. Verain MCD, Snoek HM, Onwezen MC, Reinders MJ, Bouwman EP. Sustainable food choice motives: The development and cross-country validation of the Sustainable Food Choice Questionnaire (SUS-FCQ). Food Quality and Preference [Internet] 2021 [cited 2022 Jun 10];93:104267. Available from: https://www.sciencedirect.com/science/article/pii/S0950329321001506
- 63. Brain K, Burrows TL, Rollo ME, Hayes C, Hodson FJ, Collins CE. The Effect of a Pilot Dietary Intervention on Pain Outcomes in Patients Attending a Tertiary Pain Service. Nutrients [Internet] Multidisciplinary Digital Publishing Institute; 2019 [cited 2022 Jun 8];11:181. Available from: https://www.mdpi.com/2072-6643/11/1/181

- 64. DOF Diario Oficial de la Federación [Internet]. [cited 2022 Jun 8]. Available from: https://www.dof.gob.mx/nota\_detalle.php?codigo=5259329&fecha=13/07/2012#gsc.tab=0
- 65. NORMA Oficial Mexicana NOM-015-SSA2-2010, Para la prevención, tratamiento y control de la diabetes mellitus [Internet]. [cited 2022 Jun 8]. Available from: https://www.dof.gob.mx/normasOficiales/4215/salud/salud.htm
- 66. Hickl O, Heintz-Buschart A, Trautwein-Schult A, Hercog R, Bork P, Wilmes P, Becher D. Sample Preservation and Storage Significantly Impact Taxonomic and Functional Profiles in Metaproteomics Studies of the Human Gut Microbiome. Microorganisms 2019;7:E367.
- 67. Rinninella E, Cintoni M, Raoul P, Lopetuso LR, Scaldaferri F, Pulcini G, Miggiano GAD, Gasbarrini A, Mele MC. Food Components and Dietary Habits: Keys for a Healthy Gut Microbiota Composition. Nutrients 2019;11:E2393.
- 68. Bacchetti De Gregoris T, Aldred N, Clare AS, Burgess JG. Improvement of phylum- and class-specific primers for real-time PCR quantification of bacterial taxa. Journal of Microbiological Methods [Internet] 2011 [cited 2022 Jun 10];86:351–6. Available from: https://www.sciencedirect.com/science/article/pii/S0167701211002247
- 69. Senghor B, Sokhna C, Ruimy R, Lagier J-C. Gut microbiota diversity according to dietary habits and geographical provenance. Human Microbiome Journal [Internet] 2018 [cited 2022 Jun 7];7–8:1–9. Available from: https://www.sciencedirect.com/science/article/pii/S2452231717300143
- 70. Avila-Nava A, Noriega LG, Tovar AR, Granados O, Perez-Cruz C, Pedraza-Chaverri J, Torres N. Food combination based on a pre-hispanic Mexican diet decreases metabolic and cognitive abnormalities and gut microbiota dysbiosis caused by a sucrose-enriched high-fat diet in rats. Mol Nutr Food Res 2017;61.
- 71. Meslier V, Laiola M, Roager HM, De Filippis F, Roume H, Quinquis B, Giacco R, Mennella I, Ferracane R, Pons N, et al. Mediterranean diet intervention in overweight and obese subjects lowers plasma cholesterol and causes changes in the gut microbiome and metabolome independently of energy intake. Gut 2020;69:1258–68.
- 72. Verhoog S, Taneri PE, Roa Díaz ZM, Marques-Vidal P, Troup JP, Bally L, Franco OH, Glisic M, Muka T. Dietary Factors and Modulation of Bacteria Strains of Akkermansia muciniphila and Faecalibacterium prausnitzii: A Systematic Review. Nutrients 2019;11:E1565.
- 73. Ramirez-Farias C, Slezak K, Fuller Z, Duncan A, Holtrop G, Louis P. Effect of inulin on the human gut microbiota: stimulation of Bifidobacterium adolescentis and Faecalibacterium prausnitzii. Br J Nutr 2009;101:541–50.
- 74. Akkermansia muciniphila and improved metabolic health during a dietary intervention in obesity: relationship with gut microbiome richness and ecology | Gut [Internet]. [cited 2022 Jun 7]. Available from: https://gut.bmj.com/content/65/3/426
- 75. Scher JU, Sczesnak A, Longman RS, Segata N, Ubeda C, Bielski C, Rostron T, Cerundolo V, Pamer EG, Abramson SB, et al. Expansion of intestinal Prevotella copri correlates with enhanced susceptibility to arthritis. Elife 2013;2:e01202.
- 76. Asnicar F, Berry SE, Valdes AM, Nguyen LH, Piccinno G, Drew DA, Leeming E, Gibson R, Le Roy C, Khatib HA, et al. Microbiome connections with host metabolism and habitual diet from 1,098 deeply phenotyped individuals. Nat Med [Internet] Nature Publishing Group; 2021 [cited 2022 Jun 7];27:321–32. Available from: https://www.nature.com/articles/s41591-020-01183-8
- 77. Laue H, Smits THM, Schumacher UK, Claros MC, Hartemink R, Cook AM. Identification of Bilophila wadsworthia by specific PCR which targets the taurine:pyruvate aminotransferase gene. FEMS Microbiol Lett 2006;261:74–9.
- 78. Zinöcker MK, Lindseth IA. The Western Diet-Microbiome-Host Interaction and Its Role in Metabolic Disease. Nutrients 2018;10:E365.

- 79. Jamar G, Santamarina AB, Dias GC, Masquio DCL, de Rosso VV, Pisani LP. Relationship between fatty acids intake and Clostridium coccoides in obese individuals with metabolic syndrome. Food Res Int 2018;113:86–92.
- 80. Furet J-P, Quénée P, Tailliez P. Molecular quantification of lactic acid bacteria in fermented milk products using real-time quantitative PCR. Int J Food Microbiol 2004;97:197–207.
- 81. Gila-Díaz A, Arribas SM, López de Pablo ÁL, López-Giménez MR, Phuthong S, Ramiro-Cortijo D. Development and Validation of a Questionnaire to Assess Adherence to the Healthy Food Pyramid in Spanish Adults. Nutrients [Internet] Multidisciplinary Digital Publishing Institute; 2020 [cited 2022 Jun 8];12:1656. Available from: https://www.mdpi.com/2072-6643/12/6/1656
- 82. WMA The World Medical Association-Declaración de Helsinki de la AMM Principios éticos para las investigaciones médicas en seres humanos [Internet]. [cited 2022 Jun 8]. Available from: https://www.wma.net/es/policies-post/declaracion-de-helsinki-de-la-amm-principios-eticos-para-las-investigaciones-medicas-en-seres-humanos/
- 83. Reglamento de la Ley General de Salud en Materia de Investigación para la Salud. :31.
- 84. Ley Federal de Protección de Datos Personales en Posesión de los Particulares. :18.
- 85. Salud S de. RECOMENDACIONES PARA PERSONAL DE SALUD [Internet]. gob.mx. [cited 2022 Jun 8]. Available from: http://www.gob.mx/salud/documentos/informacion-para-personal-de-salud

## **Supplementary Material**

Supplementary Material 1. Token economy system cut-off points

Table SM1.1. Scores according to the frequency of physical activity according to the type of activity

| Physical activity | Frequency for obtaining points | Score |
|---|---|---|
| Cardiovascular exercises (any | Once a week | 1 |
| including Walking, Jogging, | 2 times a week | 2 |
| Running, Aerobics, Zumba or | 3 times a week | 3 |
| dance, Cycling, Swimming) | 4 times a week | 4 |
| | 5 times a week | 5 |
| or | 6 times a week | 6 |
| Strength or resistance exercises — | 7 times a week | 7 |
| (any including Crossfit, Weights, Multifunctional Focused exercises (for example, sit-ups, squats, push-ups) | < once a week | 0 |
| | Once a week | 1 |
| | 2 times a week | 2 |
| | 3 times a week | 3 |
| Combination of cardio and | 4 times a week | 4 |
| strength exercises | 5 times a week | 5 |
| | 6 times a week | 6 |
| | 7 times a week | 7 |
| | < once a week | 0 |

Table SM1.2. Scores according to duration and intensity according to the type of physical activity

| Туре | Duration | Intensity | Score |
|---|---|---|---|
| | Less than 10 minutes | Mild | 0.5 |
| | 10 to 29 minutes | Mild | 1 |
| | 30 to 59 minutes | Mild | 2 |
| C 1' 1 | 60 to 120 minutes | Mild | 3 |
| Cardiovascular | More than 120 minutes, but | Mild | 4 |
| exercises (any | less than 240 minutes | | |
| including Walking, | More than 240 minutes | Mild | 4 points and send a message not |
| Jogging, Running,<br>Aerobics, Zumba or | | | to exceed the amount of exercise |
| dance, Cycling, | Less than 10 minutes | Moderate | 1 |
| Swimming) | 10 to 29 minutes | Moderate | 2 |
| 5 willining) | 30 to 59 minutes | Moderate | |
| or | 60 to 120 minutes | Moderate | 6 |
| 01 | More than 120 minutes, but | Moderate | 8 |
| Strength or resistance | less than 240 minutes | Moderate | o o |
| exercises (any | More than 240 minutes | Moderate | 8 points and send a message not |
| including Crossfit, | Wiore than 240 influtes | Moderate | to exceed the amount of exercise |
| Weights, | Less than 10 minutes | Intense | 2 |
| Multifunctional | 10 to 29 minutes | Intense | 4 |
| Focused exercises | 30 to 59 minutes | | 8 |
| (for example, sit-ups, | | Intense | <u> </u> |
| squats, push-ups) | 60 to 120 minutes | Intense | |
| | More than 120 minutes, but less than 240 minutes | Intense | 16 |
| | More than 240 minutes | т., | 16 1 1 1 |
| | More than 240 minutes | Intense | 16 points and send a message not to exceed the amount of exercise |
| | Logg than 10 minutes of each | Mild | to exceed the amount of exercise |
| | Less than 10 minutes of each 10 to 29 minutes of each | | 2 |
| | | Mild | 2 |
| | 30 to 59 minutes of each | Mild | 4 |
| | 60 to 120 minutes of each | Mild | 6 |
| | More than 120 minutes, but | Mild | 8 |
| | less than 240 minutes of each | 3 6'1 1 | |
| | More than 240 minutes of | Mild | 8 points and send a message not |
| | each | | to exceed the amount of exercise |
| | Less than 10 minutes of each | Moderate | 2 |
| | 10 to 29 minutes of each | Moderate | 4 |
| Combination of | 30 to 59 minutes of each | Moderate | 6 |
| cardio and strength | 60 to 120 minutes of each | Moderate | 8 |
| exercises | More than 120 minutes, but | Moderate | 10 |
| 0.1010100 | less than 240 minutes of each | | |
| | More than 240 minutes of | Moderate | 8 points and send a message not |
| | each | | to exceed the amount of exercise |
| | Less than 10 minutes of each | Intense | 4 |
| | 10 to 29 minutes of each | Intense | 8 |
| | 30 to 59 minutes of each | Intense | 16 |
| | 60 to 120 minutes of each | Intense | 24 |
| | More than 120 minutes, but | Intense | 32 |
| | More than 120 minutes, but less than 240 minutes of each | Intense | 32 |
| | More than 120 minutes, but<br>less than 240 minutes of each<br>More than 240 minutes of | Intense | 32 points and send a message not |

Table SM1.3. Scores according to the frequency of food consumption by groups

| Food group | Points for consumption frequency | Score |
|---|---|---|
| | Once a week | 1 |
| | 2 times a week | 2 |
| | 3 times a week | 3 |
| Mexican food and dishes | 4 times a week | 4 |
| Mexican food and dishes | 5 times a week | 5 |
| | 6 times a week | 6 |
| | 7 times a week | 7 |
| | < once a week | 0 |
| | Once a week | 1 |
| | 2 times a week | 0 |
| | 3 times a week | 0 |
| Mexican desserts and drinks | 4 times a week | 0 |
| | 5 times a week | 0 |
| | 6 times a week | 0 |
| | 7 times a week | 0 |
| | Once a week | 1 |
| | 2 times a week | 2 |
| | 3 times a week | 3 |
| Fruits, vegetables, legumes, dairy, | 4 times a week | 4 |
| seeds and healthy fats, eggs | 5 times a week | 5 |
| | 6 times a week | 6 |
| | 7 times a week | 7 |
| | < once a week | 0 |
| | Once a week | 3 |
| | 2 times a week | 2 |
| | 3 times a week | 1 |
| Fish and shellfish, chicken and other | 4 times a week | 0 |
| white meats — | 5 times a week | 0 |
| | 6 times a week | 0 |
| | 7 times a week | 0 |
| | 0 times a week | 7 |
| | Once a week | 1 |
| | 2 times a week | 0 |
| Red and processed meats, Ultra- | 3 times a week | 0 |
| processed foods, Foods high in sugars, — trans and saturated fats — | 4 times a week | 0 |
| trans and saturated fats | 5 times a week | 0 |
| | 6 times a week | 0 |
| | 7 times a week | 0 |

Table SM1.4. Scores by frequency of consumption

| Food group | Consumption quantities | Score |
|---|---|---|
| M : C 1 11:1 | < recommended portion or > minimum portion | 1 |
| Mexican foods and dishes, | Recommended portion | 2 |
| fruits, vegetables, legumes, dairy products, seeds and | < recommended maximum or > recommended portion | 1 |
| healthy fats, eggs | > the recommended maximum or < the recommended minimum | 0 |
| Fish and shellfish, chicken | Minimum portion | 3 |
| and other white meats, Red | < Recommended portion > minimum portion | 2 |
| and processed meats, Ultra- | > recommended portion < maximum portion | 1 |
| processed foods, Foods high<br>in sugars, trans and saturated<br>fats | > Maximum portion | -1 |

Note: recommend amount of consumption will be determined by the linear optimization programing. An example is shown in Table SM1.5.

Table SM1.5. Examples of recommended amounts of consumption by food groups including the target foods of the intervention

| | | | Examples of a | mounts of consum | otion |
|---|---|---|---|---|---|
| Consumption | option Group by Food objective | | Average<br>Recommended Serving | Ran | ge |
| | | | | Minimum | Maximum |
| | | Chilaquiles with or without egg and/or chicken | 1 cup (160 g) | 80 g | 240 g |
| | | Mexican style egg (tomato, onion, chili, nopal) | 1 plate (220 g) | 110 g | 330 g |
| | | Quesadilla of corn tortilla (without meat) | 1 piece (60 g) | 30 g | 90 g |
| | | Beans taco | 1 piece (60 g) | 30 g | 90 g |
| | | Panela cheese and beans torta (not meat) | 1 piece (197 g) | 98.5 | 295.5 g |
| | | Chicken tamal (no red meat) | 1 piece (200 g) | 100 g | 300 g |
| | | Tamal of ash, chard, or cheese (without red meat) | 1 piece (200 g) | 100 g | 300 g |
| Daily (at least | | Sweet tamal (corn, fruits) | 1 piece (172 g) | 86 g | 258 g |
| 1 food from | | Mole with chicken | 1 plate (334 g) | 167 g | 501 g |
| the group) | | Chicken or vegetarian (mushroom) pozole | 1 plate (300 g) | 150 g | 450 g |
| | | Chicken or cheese flute (no red meat) | 1 piece (75 g) | 37.5 g | 112.5 g |
| | | Bean or chicken sope (no red meat) | 1 piece (75 g) | 37.5 g | 112.5 g |
| | Mexican food | Chicken or cheese enchilada (no red meat) | 1 piece (75 g) | 196.5 g | 589.5 g |
| | and dishes | Fish or chicken taco (no beef or pork) | 1 piece (75 g) | 37.5 g | 112.5 g |
| | | Bean burrito (no meat) | 1 piece (100 g) | 50 g | 150 g |
| | | Fresh water without sugar | 1 cup (240 ml) | 120 ml | 360 ml |
| | | Toast with beans or chicken | 1 big toast (174 g) | 87 g | 261 g |
| | | Rice pudding | ½ cup (178 g) | 89 g | 267 g |
| | | Flan | 1 piece (120 ml) | 60 ml | 180 ml |
| | | Capirotada | 1 slice (60 g) | 30 g | 90 g |
| 1 4 | | Sweet bread | 1 piece (63 g) | 31.5 g | 94.5 g |
| 1 time per | | Atole in water | 1 cup (240 ml) | 120 ml | 360 ml |
| week | | Atole in milk or champurrado | 1 cup (240 ml) | 120 ml | 360 ml |
| | | Tejuino | 2 cups (418 ml) | 209 ml | 627 ml |
| | | Tuba | 1 cup (240 ml) | 120 ml | 360 ml |
| | _ | Tepache or honey water | 1 cup (240 ml) | 120 ml | 360 ml |

Table SM1.5. Continuation: Examples of recommended amounts of consumption by food groups including the target foods of the intervention

| Examples of amounts of consumption | | | | ption | |
|---|---|---|---|---|---|
| Consumption | Group by | Food | Average | Ran | ge |
| | objective | | Recommended Serving | | |
| | | Papaya | 1 cup (140 g) | 70 g | 210 g |
| | | Tuna | 1 piece (70 g) | 35 g | 105 g |
| | | Pineapple | 1 cup (165 g) | 82.5 g | 247.5 g |
| Daily (at least | | Soursop | ½ piece (175 g) | 87.5 g | 262.5 g |
| 1 food from | Fruits | Guava | 2 pieces (83 g) | 41.5 g | 124.5 g |
| the group) | | Capulín | 1 cup (32 g) | 16 g | 48 g |
| | | Pitaya | 1 piece (50 g) | 25 g | 75 g |
| | | Nance | 5 pieces (15 g) | 7.5 g | 22.5 g |
| | | Creole plum | 2 pieces (105 g) | 52.5 g | 157.5 g |
| | | Zucchini | 1 piece (91 g) | 45.5 g | 136.5 g |
| | | Pumpkin | ½ cup (110 g) | 55 g | 165 g |
| | | Onion | ½ cup (58 g) | 29 g | 87 g |
| | | Mushrooms | 1 cup (93 g) | 46.5 g | 139.5 g |
| | | Chayote | ½ cup (80 g) | 40 g | 120 g |
| Dailer (at 1 a a t | | Spicy chili | 1 cup (30 g) | 15 g | 45 g |
| Daily (at least 1 food from | Vegetables ——— | Huitlacoche | 1/3 cup (66 g) | 33 g | 99 g |
| the group) | vegetables | Tomato | 2 pieces (124 g) | 62 g | 186 g |
| the group) | | Nopales | 2 pieces (134 g) | 67 g | 201 g |
| | | Bell pepper | 1 piece (64 g) | 32 g | 96 g |
| | | Poblano chili | 1/2 piece (32 g) | 16 g | 48 g |
| | | Quelites | ½ cup (66 g) | 33 g | 99 g |
| | | Green tomato | 5 pieces (86 g) | 43 g | 129 g |
| | | Purslane | 1 cup (115 g) | 57.5 g | 172.5 g |
| | | Corn tortilla | 1 piece (30 g) | 15 g | 45 g |
| Dailer (at 1 a a t | | Baked corn toast | 2 pieces (20 g) | 10 g | 30 g |
| Daily (at least 1 food from | Whole grains - | Corn dough | 1 ball (45 g) | 22.5 g | 67.5 g |
| the group) | Whole grains | Unsweetened amaranth | ½ cup (16 g) | 8 g | 24 g |
| me group) | | Sweetened amaranth | <sup>1</sup> / <sub>4</sub> cup (16 g) | 8 g | 24 g |
| | | Sweet potato | 1/3 cup (69 g) | 34.5 g | 103.5 g |

Table SM1.5. Continuation: Examples of recommended amounts of consumption by food groups including the target foods of the intervention

| Examples of amounts of consumpti | | | otion | | |
|---|---|---|---|---|---|
| Consumption | Group by objective | · | | Average Range ecommended Serving | |
| | | Pot beans | ½ cup (86 g) | 43 g | 129 g |
| Daily (at least | | Fried beans | 1/3 cup (75 g) | 37.5 g | 112.5 g |
| 1 food from | Legumes | Cooked lentils | ½ cup (99 g) | 49.5 g | 148.5 g |
| the group) | | Cooked chickpeas | ½ cup (82 g) | 41 g | 123 g |
| | | Baked beans | ½ cup (85 g) | 42.5 g | 127.5 g |
| | | Curd | 3 tablespoons (36 g) | 18 g | 54 g |
| | | Fresh cheese | 1 slice (40 g) | 20 g | 60 g |
| Daily (at least | | Panela cheese | 1 slice (40 g) | 20 g | 60 g |
| 1 food from | Dairy products | Natural yogurt | 1 cup (227 g) | 113.5 g | 340.5 |
| the group) | | Whole milk | 1 cup (240 ml) | 120 ml | 360 ml |
| | | Semi-skimmed milk | 1 cup (240 ml) | 120 ml | 360 ml |
| | | Skim milk (light) | 1 cup (240 ml) | 120 ml | 360 ml |
| | | Avocado | 1/3 piece (31 g) | 15.5 g | 46.5 g |
| Dailer (at 1aaat | | Dried beans | <sup>1</sup> / <sub>4</sub> cup (38 g) | 19 g | 57 g |
| Daily (at least 1 food from | Seeds and | Pumpkin seeds | 2 tablespoons (15 g) | 7.5 g | 22.5 g |
| the group) | healthy fats | Chia seeds | 5 teaspoons (12 g) | 6 g | 18 g |
| the group) | | Peanuts | 14 pieces (12 g) | 6 g | 18 g |
| | | Canola oil | 1 teaspoon (5 g) | 5 ml | 15 ml |
| Daily (at least | | Complete chicken egg | 1 piece (44 g) | 22 g | 66 g |
| 1 food from the group) | Eggs | Egg white | 2 pieces (66 g) | 33 g | 99 g |
| 0 4 2 4 3 | Piul 1 | White fish | 1 portion (40 g) | 0 g | 60 g |
| 0 to 3 times a | Fish and ——————————————————————————————————— | Octopus | 1 portion (25 g) | 0 g | 37.5 g |
| week | SHCHIISH | River prawn | 4 pieces (110 g) | 0 g | 165 g |
| 0 to 3 times a | Chicken and | Grilled chicken | 1 portion (29 g) | 0 g | 58 g |
| | other white | Chicken in piece | 1/3 piece (29 g) | 0 g | 58 g |
| week | meat | Insects (maguey worms, crickets) | 1 portion (35 g) | 0 g | 52.5 g |

Table SM1.5. Continuation: Examples of recommended amounts of consumption by food groups including the target foods of the intervention

| | | | Examples of an | nounts of consum | ption |
|---|---|---|---|---|---|
| Consumption | Group by objective | Food | Average<br>Recommended Serving | Ran | ge |
| | <b>V</b> | Beef | 1 portion (14 g) | 0 g | 60 g |
| | | Pork Meat | 1 portion (14 g) | 0 g | 60 g |
| | | Rabbit | 1 portion (29 g) | 0 g | 58 g |
| | | Pork or turkey ham | 1 slice (10.5 g) | 0 g | 21 g |
| | | Pork or turkey sausage | 1 slice (14 g) | 0 g | 60 g |
| | | Longaniza, chorizo, pepperoni or salami | 1 portion (14 g) | 0 g | 30 g |
| | | Beef or pork tacos | 1 piece (75 g) | 0 g | 112.5 g |
| | | Quesadilla with meat, gringa or synchronized (with sausages | 1 piece (60 g) | 0 g | 90 g |
| | | or meats) | | _ | |
| 0 to 1 time a | Red and | Enchilada with beef or pork | 1 piece (75 g) | 0 g | 112.5 g |
| week | processed meats | Flute with beef or pork | 1 piece (75 g) | 0 g | 112.5 g |
| | | Sope with beef or pork | 1 piece (75 g) | 0 g | 112.5 g |
| | | Pork pozole | 1 plate (300 g) | 0 g | 450 g |
| | | Offal | 1 plate (300 g) | 0 g | 450 g |
| | | Birria | 1 plate (200 g) | | |
| | | Meat tamal | 1 piece (200 g) | 0 g | 300 g |
| | | Torta (marinated, meat, drowned) | 1 piece (197 g) | 0 g | 295.5 g |
| | | Beef burrito | 1 piece (100 g) | 0 g | 150 g |
| | | Toast with beef or pork | 1 large piece of toast<br>(174 g) | 0 g | 261 g |
| | | Soft drink with sugar | <sup>1</sup> / <sub>4</sub> can (92 ml) | 0 ml | 138 ml |
| | | Sugar free soft drink | <sup>1</sup> / <sub>4</sub> can (92 ml) | 0 ml | 138 ml |
| | | Packaged juice | 1/3 cup (80 ml) | 0 ml | 120 ml |
| 0 to 1 time a | Ultra-processed | Packaged cookies | 1 piece (10.5 g) | 0 g | 15.75 g |
| week | foods | Box cereals | ½ cup (16 g) | 0 g | 24 g |
| | | Instant soup | 1 piece (64 g) | 0 g | 96 g |
| | | Packaged cupcakes (pingüinos, chocorroles, gansitos) | 1/2 piece (25 g) | 0 g | 37.5 g |
| | | Packaged potato chips or snacks | 6 piece (18 g) | 0 g | 27 g |

Table SM1.5. Continuation: Examples of recommended amounts of consumption by food groups including the target foods of the intervention

| | | | Examples of an | nounts of consum | ption |
|---|---|---|---|---|---|
| Consumption | Group by | | | Rar | nge |
| | objective | | Recommended Serving | | |
| | | Table sugar to sweeten | 1 teaspoon (4 g) | 0 g | 6 g |
| | | Fresh water with sugar | 1 cup (240 ml) | 0 g | 360 ml |
| | | Industrialized jams | 1 tablespoon (17 g) | 0 g | 25.5 g |
| 0 . 1 .: | г 11'1' | Industrialized syrups and honeys | 1 teaspoon (7 g) | 0 g | 10.5 g |
| | Foods high in added and free | Cake or pie (thin slice) | 1 slice (28 g) | 0 g | 32 g |
| 0 to 1 time a week | | Vegetable oil (not olive or canola) | 1 teaspoon (5 ml) | 0 g | 7.5 ml |
| WEEK | sugars, trans and ——————————————————————————————————— | Salt added to already prepared foods | 1 pinch (2 g) | 0 g | 3 g |
| | Saturated rats | Vegetable shortening | 1 teaspoon (5 g) | 0 g | 7.5 g |
| | | Margarine | 1 teaspoon (5 g) | 0 g | 7.5 g |
| | | | Lard | 1 teaspoon (5 g) | 0 g |
| | | Butter | 1 teaspoon (5 g) | 0 g | 7.5 g |

Supplementary Material 2. Inclusion, exclusion, and elimination criteria

Table SM2.1. Inclusion, exclusion, and elimination criteria

| | Study Criteria | |
|---|---|---|
| Inclusion | Exclusion | Elimination |
| Being between 18 and 35 years old | Not signing the informed consent | Not completing the questionnaires |
| Being Mexican | Not accepting to donate blood and/or stool samples | Do not allow the extraction of blood and / or delivery of stool sample |
| Reside in the South of Jalisco for at least 1 year | Not being able to stand up to take anthropometric data | Failure to complete the 7-week intervention or 7-week follow-up |
| Levels of physical activity<br>below what is recommended<br>and what is established as a<br>criterion for inclusion in the<br>study (Table SM2) | Perform levels of physical activity above the minimum established as criteria for inclusion in the study (Table SM2) | |
| Consuming amounts of food<br>below or above that<br>established as criteria for<br>inclusion in the study or in a<br>lesser or greater frequency<br>than recommended, according<br>to the type of food (Table<br>SM2) | Consume adequate levels of the foods to be promoted in the intervention program (Table SM2) | |
| Have a Smartphone | Being pregnant or lactating | |
| Not having consumed antibiotics at least 3 months before the intervention | Suffer from a chronic disease<br>such as type 2 diabetes mellitus,<br>arterial hypertension,<br>dyslipidemia, under medication | |
| Have a BMI between 18.5 and 40 | Suffering from an autoimmune disease such as type 1 diabetes, hypo or hyperthyroidism | |
| Not having a medical diagnosis of chronic disease under pharmacological treatment | Having a gastrointestinal disease such as Crohn's disease, ulcerative colitis, etc. | |
| Not having a medical diagnosis of gastrointestinal disease | Having used antibiotics less than 3 months ago | |
| | Taking antidepressant medications or corticosteroids | |
| | Consume probiotics or nutritional supplements, except protein | |
| | powder | |

Table SM2.2 Cut-off points to establish inadequate consumption and physical activity, to be included in the research

| Physical activity | Inclusion criteria | |
|---|---|---|
| Type of physical activity | | Light |
| Weekly frequency | < 3 tir | nes per week |
| Minutes per day | < 30 m | inutes per day |
| Earl amount | Consumption to be | Frequency of consumption to |
| Food group | included in the study | be included in the study |
| Mexican food and dishes | $< 100 \text{ g p}^{-1} \text{d}^{-1}$ | < 7 times a week |
| Fruits | $< 400 \text{ g p}^{-1} \text{d}^{-1}$ | < 7 times a week |
| Vegetables | $< 400 \text{ g p}^{-1} \text{d}^{-1}$ | < 7 times a week |
| Whole cereals | $< 200 \text{ g p}^{-1} \text{d}^{-1}$ | < 7 times a week |
| Legumes | $< 60 \text{ g p}^{-1} \text{d}^{-1}$ | < 7 times a week |
| Seeds and healthy fats | $< 80 \text{ g p}^{-1} \text{d}^{-1}$ | < 7 times a week |
| Dairy products | $> 250 \text{ ml p}^{-1}\text{d}^{-1}$ | > 5 times a week |
| Eggs | $> 25 \text{ g p}^{-1} \text{d}^{-1}$ | > 5 times a week |
| Fish and shellfish | $> 28 \text{ g p}^{-1} \text{d}^{-1}$ | > 3 times a week |
| Chicken | $> 29 \text{ g p}^{-1} \text{d}^{-1}$ | > 3 times a week |
| Red and processed meats | $> 7 \text{ g p}^{-1} \text{d}^{-1}$ | > once a week |
| Ultra-processed foods | $> 10 \text{ g p}^{-1} \text{d}^{-1}$ | > once a week |
| Added and free sugars and foods high in | $> 31 \text{ g p}^{-1} \text{d}^{-1}$ | > once a week |
| trans and saturated fats | | |

# Supplementary Material 3. Clinical history which will be uploaded to the mobile application

Table SM3.1 Initial Assessment Questionnaire

| | | | Clinic history | |
|---|---|---|---|---|
| | | | l and sociodemographic data | |
| Last name: Middle name: | | | Name: | |
| Cell phone: | | | Email: | |
| Age: | | | Date of Birth: | |
| Sex: | | | Country of birth: | |
| City of residence: | | | State of birth: | |
| Time living there: | | | Occupation | |
| Less than 1 month | | | Officer, director or boss | |
| 1 to 6 months | | | Professional or technician | |
| 6 to 12 months | | | Auxiliary worker in administrative activities | |
| 1 to 3 years | | | Merchant, sales clerk, or sales agent | |
| 3 to 6 years | | | Workers in personal and surveillance services | |
| 6 to 9 years | | | Worker in agricultural, livestock, forestry, hunting or fishing activities | |
| 10 years or more | | | Craft worker | |
| Lifetime | | | Industrial machinery operator, assemblers, chauffeur or transport driver | |
| Lifetime | | | Workers in elementary and support activities | |
| , | 744: | | | d support activities |
| | Education | | Student | |
| Did not sudy | | | Unemployed | |
| Unfinished primary | | | Retired | |
| Finished elementary school | | | Other (specify): | |
| Unfinished high school | | | Days a week that work | |
| High school finished | | | 1 | |
| Unfinished high school | | | 2 | |
| School completed | | | 3 | |
| Unfinished technical career | | | 4 | |
| Technical career finished | | | 5 | |
| Undergraduate student | | | 6 | |
| Unfinished degree | | | 7 | |
| Completed bachelor's degree | | | Modality | |
| Master's degree | | | Face-to-face | |
| Doctorate Doctorate | | | Online | |
| | | | Mixed | |
| Other: | Specialty Others | | | Online until further notice |
| | | 11 | | |
| Individual and family Individual expenditure on food per month | | | sehold expenditure on food reeding (MXN pesos) | |
| month MXN) | (MXN pesos) | | | |
| -0 - 2,699 | | | 0 – 500 | Favorite foods |
| 2,7–0 - 6,799 | -0 - 200 | | 500 – 1,000 | |
| 6,8–0 - 11,599 | 2-0 - 500 | | 1,000 – 3,000 | Foods you don't like |
| 11,6–0 - 34,999 | 500 – 800 | | 3,000 – 6,000 | |
| 35,000 - 84,999 | 800 – 1,000 | | 6,000 – 9,000 | Food allergies and intolerances |
| + 85,000 | 1,500- 2,000 | | 10,0-0 - 13,000 | Lactose |
| , i | 2,500 – 3,000 | | 13,000 - 16,000 | Seafood |
| | 3,000 – 3,500 | | 16.000 - 20.000 | Gluten |
| | + 4.000 | | + 20.000 | Fresas |
| | Diet and physical activity | tv | . 20,000 | Nuts |
| Main place of food | Who cooks the food you | | Are you currently | Peanuts |
| | Who cooks the food you | · Cat: | 0.11 | 1 Canata |
| Tionguis | Ma | | following a specific diet? | Othors (amosify) |
| Tianguis | Me | - | | Others (specify): |
| Market | Mother | - | Yes | |
| Retail supermarket<br>(Soriana, Walmart) | Father | | To lose weight | |
| Wholesale | Economic Kitchen | | To gain weight | |
| supermarket (Sam's,<br>Costco) | Establish Hamila | Leonomic Kitchen | | To game in origin |
| Butcher shop | Restaurants | Pastaurants | | Ketogenic |
| · | | | | |
| Creamery | | | Vegetarian (ovo-lacto, ovo or lacto) | |
| Fruit store Others (specify): | | | Intermittent fasting | |
| Others (specify): | | | Vegan | |
| | | | Mediterranean | |
| | | | DASH or diet to stop hype<br>Others (specify): | ertension |

Table SM3.1 Continuation: Initial Assessment Questionnaire

| | | Clinic history | |
|---|---|---|---|
| Cumuntly daing physical and | iia. | Physical activity | Type of activity |
| Currently doing physical act | 11VITY | | Type of activity Walking |
| Less than 3 times a week | | | warking |
| | activity of at least 20 minutes per da | Jogging | |
| | to vigorous activity or walking at le | | Run |
| | ous activity for at least 60 minutes a | Aerobics, Zumba or dance | |
| | o vigorous activity or even walking | Cycling | |
| Times a week | Type of activity | Minutes a day | Swimming |
| 1 | | 10 | Crossfit |
| 2 | | 20 | Weightlifting |
| 3 | | 30 | Multifunctional |
| 4 | | 40 | Focused exercises (write |
| | | | which ones, e.g. sit-ups, sit- |
| | | | ups, push-ups) |
| 5 | | 50 | Other: |
| 6 | | 60 | |
| 7 | | 90 | <del> </del> |
| | Intensity | 120 | <del> </del> |
| Mild | | 150 | <del> </del> |
| Moderate | | 180 | <del> </del> |
| Intense | | 210 | |
| | | 240 or more | |
| | | Other: | |
| | | Anthropometric data | |
| Estimated weight for you: | | Size in centimeters | |
| ** * 1 . / | | estimated by you: | 77.0 |
| Height (centimeters): | | Weight (kg): | BMI: |
| Fat percentage: | | Muscle mass: | Body water: |
| Metabolic age: | | Metabolic rate: | Visceral fat: |
| Waist circumference: | D' 1 ' 1' 1' 4 | Hip circumference: | Bone mass: |
| Etinlu | Biochemical indicators | | Clinical indicators |
| Fasting glucose Glucose 2 hours after eating | | | Blood pressure Acanthosis nigricans |
| | | | Signs and symptoms of nutritional deficience |
| Triglycerides Total cholesterol | | | Overall status |
| LDL cholesterol | | | Very tired |
| HDL cholesterol | | | Dizziness |
| Gut microbiota | | | Very thirsty |
| Gut inicionota | Gastrointestinal signs and sympto | ims | Frequent urination |
| Abdominal swelling | Gastromestmar signs and sympto | inis | Very hungry |
| How often does it happen? | | | Do your feet or hands swell? |
| Diarrhea | | | What time of day does it occur? |
| How often does it happen? | | | How often does it happen? |
| Constipation | | | How many hours do you spend |
| Consequence | | | sitting a day? |
| How often does it happen? | | | How many hours do you spend |
| | | | standing a day? |
| Reflux | | | Nose bleed |
| How often does it happen? | | | How often does it happen? |
| Abdominal swelling | | | Red spots on your skin or bruises |
| | | | for no reason |
| How often does it happen? | | | How often does it happen? |
| | Nails | | Hair |
| Brittle nails | | Hair loss | |
| Have you recently performe | d any cosmetic treatment on your na | ails? Brittle hair Is your hair | dyed or undergoing any cosmetic |
| | | treatment? | |
Table SM3.1 Continuation: Initial Assessment Questionnaire

| Clinic history | | |
|---|---|---|
| Signs and symptoms of nutritional d | leficiencies | |
| Mouth | Sueño | |
| Cuts at the corners of your mouth | How many hours do you sleep a day? | |
| How often does it happen? | Do you rest at night? | |
| Tongue swelling | Do you wake up during the night? | |
| How often does it happen? | How often does it happen? | |
| Gum inflammation | How many hours do you sleep a day? | |
| How often does it happen? | Do you rest at day? | |
| Solar exposition | | |
| How many minutes do you expose yourself to the sun per day? | Do you cover your skin with long-sleeved cl<br>pants, a cap or a hat? | lothing, |
| Less than 5 minutes | Always | |
| 5 to 10 minutes | Sometimes | |
| 10 to 15 minutes | Never | |
| 15 to 20 minutes | Do you use sunscreen? | |
| 20 to 30 minutes | Yes | |
| 30 minutes to 1 hour | No | |
| More than 1 hour | How many days do you expose yourself | |
| | to the sun per week? | |
| Type of delivery | 1 | |
| You were born for: | 2 | |
| Vaginal delivery | 3 | |
| Caesarean section | 4 | |
| Notes: | 5 | |
| | 6 | |
| | 7 | |
| Lactation | Write for how long | |
| Exclusive breastfeeding | | |
| Formula feeding (if you received only artificial milk as food) | Observations: | |
| Mixed breastfeeding (if in addition to breastfeeding you received any artificial milk) | | |
| Supplemented breastfeeding (if non-dairy solid or liquid foods were received in addition to breastfeeding) | | |
| Mixed supplemented breastfeeding (if it was a breastfed infant, who also | | |
| received some artificial milk and solid or liquid foods) | | |
| Complemented artificial feeding (if when breastfeeding you received artificial milk and solid or liquid foods) | | |
| Festivities | | |
| Please write the main holidays you celebrate and on the right side wr | ite the main foods you eat on these holidays | |
| Festivity | Food eaten on the holiday | |
| restivity | rood eaten on the honday | |
| _ YY - 1 | | |
| Hygiene habits | | |
| How often do you take a bath? | | |
| How many times do you brush your teeth a day? | | |
| Is the street where you live paved? | | |
| What type of flooring does your house have? | | |
| Do you have pets? What type? | | |

Table SM3.1 Continuation: Initial Assessment Questionnaire

| | Per | sonal ar | nd fami | ly histo | rv | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | ny dise | | | | | | | | | |
| Mark pathology | | | | | | | | | | | | | |
| | | | | | | | | | | suc | | | |
| | | l ä | es | | | | | | w . | ficie | | | |
| | | nsic | erid | _ | | | | g | l iriti | Insi | | | |
| | stes | erte | lyc | ero | it: | | lism | disr | art | .E | b | | |
| | iabe | hyp | tri. | lest | col | | roic | /roi | oid | Leng | eas | on | |
| | 2 d | ial ] | ıted | chc | sno | is . | thy | l thy | mat | nic | dis | essi | |
| | Type 2 diabetes | Arterial hypertension | Elevated triglycerides | High cholesterol | Nervous colitis | Cancer | Hypothyroidism | Hyperthyroidism | Rheumatoid arthritis | Chronic renal insufficiency | Heart disease | Depression | Other |
| | <u> </u> | < | Ш | Η | Z | O | 田 | <sup>II</sup> | ~ | O | H | | 0 |
| If you selected the other option, specify which or which | | | | | | | | | | | | | |
| | one in | | | ffon fr | ant- | ligang - 9 | | | | | | | |
| Does any Father | one in | your iai | iiiiy su | iter iro | in any c | usease? | | | | | | | |
| Mother | | | | | | | | | | | | | |
| Brother | | | | | | | | | | | | | |
| Sister | | | | | | | | | | | | | |
| Paternal grandfather | | | | | | | | | | | | | |
| Paternal grandmother Maternal grandfather | | | | | | | | | | | | | |
| Maternal grandmother | | | | | | | | | | | | | |
| Paternal uncle | | | | | | | | | | | | | |
| Paternal aunt | | | | | | | | | | | | | |
| Maternal uncle | | | | | | | | | | | | | |
| Maternal aunt | | | | | | | | | | | | | |
| Other: Do you curre | ntly tol | co onti | madiant | ions on | d/or su | nnlamai | atc? | | | | | | |
| Medicines Bo you curr | litiy tai | ally I | licuicai | 10115 411 | u/or su | ppiemei | 115: | | | | | | |
| | | | | cin. | Clarithromycin | | | Levothyroxine | | | မ | | |
| | Ampicillin | Bezafibrate | Cephalexin | Ciprofloxacin | lom | Fluoxetine | | yro; | g g | Metformin | Omeprazole | Pravastatin | Telmisartan |
| | pici | afib | hale | rofi | ith | oxe | il. | oth | Losartan | -<br>Lou | epra | /ast | nis |
| | Am | Bez | Cep | Cip | Cla | Fluc | Insulin | Lev | Los | Met | Om | Pra | Tel |
| Other. If you selected the other option, specify which or | <u> </u> | | | | | ' ' | | ' ' | | ' ' | | ' ' | |
| which | | | | | | | | | | | | | |
| Supplements | | | | | | | | | | | | | |
| · | | | | | | | | | | | | | |
| | | | | | | | | | | | ,, | | |
| | | | | | | | | | | | -<br> rate | | |
| | nin | Д | SS | SS | C | ш | | <sub>E</sub> | m | vde | hyc | | |
| | Multivitamin | Vitamin D | Probiotics | Prebiotics | Vitamin C | Vitamin E | Iron | Calcium | Omega 3 | pov | ono | Other | |
| | -lltiv | itan | rob | rebi | itar | itar. | Ä | Calc | )me | ein | e m | Q | |
| | ₹ | > | _ <u>P</u> | Ь Р | > | > | | | | Protein powder | atin | | |
| | | | | | | | | | | _ | Creatine monohydrate | | |

Table SM3.1 Continuation: Initial Assessment Questionnaire

| | 24-hour r | eminder | |
|---|---|---|---|
| Food time | Menu / Preparation | Ingredient / Food | Quantity |
| Breakfast | | | |
| ** | | | |
| Hour: | | | |
| Place: | | | |
| Morning snack | | | |
| Hour: | | | |
| Place: | | | |
| Tiacc. | | | |
| Meal | | | |
| Hour: | | | |
| Place: | | | |
| Place: | | | |
| Ei | | | |
| Evening snack | | | |
| Hour: | | | |
| Place: | | | |
| Dinner | | | |
| Hour: | | | |
| Place: | | | |
| Milliliters of wat | er consumed throughout the day: | | |

Table SM3.1 Continuation: Initial Assessment Questionnaire

# Food frequency questionnaire

For each food, indicate how many times per month or per week you consume it. Subsequently, indicate how many times a day you consume it, the day you take it. For example, if you drink 2 cups (480 milliliters) of whole milk 3 times a week and those 3 days you drink it in the morning and at night, you drink it 3 times a week and 2 times a day, in a quantity of 2 portions. It is also important to consider the summer/winter variation. For example, if you eat ice

| tillic | s a week and those 3 days you drink it in the morning and at | cream 4 times a wee | | | | | | | | | | | | JOHSIC | iei ilie | Sulli | ilici/wi | ilitei va | папоп | . 1.01 | CXan | ipie, i | ı you c | tat ice |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Group | Food | Portion | Type, brand, flavor or preparation | *M<br>*If you<br>and go | Av<br>Iark 1<br>do no<br>to the | erage of option of consinext fo | consu<br>amo<br>ume<br>od. | ımpti<br>ong th<br>it, ch | ion l<br>iese | last y<br>3 fr<br>se th | year<br>equo<br>e op | encie<br>otion | s.<br>neve | | con<br>how<br>times<br>you<br>(C<br>option | ı do i<br>heck<br>ı per | it,<br>ny<br>y do<br>t?<br>1<br>day) | | | | | | ings | |
| | | | Тур | | nes a yea | | mo | nes a<br>onth | | | | a wee | | | | es a c | • | | Mark<br>consur | ne ea | ch ti | me yo | u eat | it) |
| | | 4 (242 ) | | Never | 1-5 | 6-11 | 1 | 2 3 | 1 | 2 | 3 | 4 5 | 6 | 7 | 1 2 | 3 | 4+ | 1/4 | 1/2 | 1 | 2 | 3 | 4 5 | 6+ |
| | 1. Whole milk | 1 cup (240 ml) | | | | | | | | | | | | _ | | | | | | | | | | |
| | 2. Semi-skim milk | 1 cup (240 ml) | | | | | _ | | _ | | _ | | | | | | | | | | | | | |
| | 3. Skim milk | 1 cup (240 ml) | | | | | | | | | | | | _ | | | | | | | | | | |
| | 4. Almond milk | 1 cup (240 ml) | | | | | _ | | _ | | _ | | | | | | | | | | | | | |
| _ | 5. Soy milk | 1 cup (240 ml) | | | | | | | | | | | | _ | | | | | | | | | | |
| Dairy | 6. Coconut milk | 1 cup (240 ml) | | | | | _ | | _ | | | | | | | | | | | | | | | |
| ã | 7. Chocolate flavored milk | 1 cup (240 ml) | | | | | | | | | | | | _ | | | | | | | | | | |
| | 8. Packaged milk shake | 1 cup (240 ml) | | | | | $\perp$ | | _ | | _ | | | | | | | | | | | | | |
| | 9. Whole yogurt (sweetened with fruit) | 1 cup (227 g) | | | | | | | | | | | | | | | | | | | | | | |
| | 10. Low-fat yogurt | 1 cup (240 g) | | | | | $\perp$ | | _ | | _ | | | | | | | | | | | | | |
| | 11. Fermented milk drink | 1 piece (80 g) | | | | | | | | | | | | _ | | | | | | | | | | |
| | 12. Bionico cream (evaporated milk with cow cream) | ½ cup (120 g) | | | | | $\perp$ | | _ | | _ | | | | | | | | | | | | | |
| | 13. Curd | 3 tablespoons (42 g) | | | | | | | | | | | | _ | | | | | | | | | | |
| , s | 14. Cottage cheese | 3 tablespoons (48 g) | | | | | ш | | ᆫ | | | | $\perp$ | | | | | | | | | | | |
| ese | 15. Fresh cheese (not in quesadillas) | 1 slice (40 g) | | | | | | | | | | | | | | | | | | | | | | |
| Cheeses | 15.1 Panela cheese (not in quesadillas) | 1slice (40 g) | | | | | ш | | ᆫ | | | | $\perp$ | | | | | | | | | | | |
| | 16. Cured cheeses consumed alone (manchego, oaxaca, asadero, mozzarella, cheddar, goat, parmesan, chihuahua), (not in quesadillas) | 1 slice (30 g) | | | | | | | | | | | | | | | | | | | | | | |
| | 17. Chicken eggs | 1 piece (60 g) | | | | | | | | | | | | | | | | | | | | | | |
| ٠ | 18. Egg white | 2 pieces (66 g) | | | | | | | | | | | | | | | | | | | | | | |
| source<br>4s | 19. Chicken with skin (chicken pieces except wings) | 1 piece (200 g) | | | | | | | | | | | | | | | | | | | | | | |
| | 20. Chicken without skin in pieces | 1 piece (200 g) | | | | | | | | | | | | | | | | | | | | | | |
| nimal | 20.1 Grilled skinless chicken fillet | 1 ration (90 g) | | | | | | | | | | | | | | | | | | | | | | |
| · Ē | 21. Turkey | 1 ration (108 g) | | | | | | | | | | | | | | | | | | | | | | |
| | 21.1 Bunny | 1 ration (90 g) | | | | | | | | | | | | | | | | | | | | | | |
| | 22. Beef steak or steak (stews, griddle) | 1 ration (90 g) | | | | | | | | | | | | | | | | | | | | | | |

| | | | <br> |
|---|---|---|---|
| | 23. Ground beef (meatballs, hash) | 1 ration (99 g) | |
| | 24. Pork (stews, grilled) | 1 ration (120 g) | |
| | 25. Sheep meat (al pastor, stews) | 1 ration (111 g) | |
| | 26. Goat meat (birria) | 1 ration (100 g) | |
| | 27. Liver or organ meats of chicken, beef or pork (brains, gizzard, heart) | 1 ration (90 g) | |
| | 28. Turkey or pork ham (besides of used in sandwich) | 1 slice (21 g) | |
| | 29. Turkey or pork sausage (other than hot dog) | 1 piece (61 g) | |
| | 30. Processed meats (pepperoni, salami, sausage, chorizo, machaca) | ½ cup (20 g) | |
| | 31. Bacon | 1 slice (16 g) | |
| | 32. Pork rinds | ½ cup (24 g) | |
| | 33. White fish (tilapia, sole) | 1 ration (120 g) | |
| | 34. Blue fish (salmon, tuna, red snapper) | 1 ration (120 g) | |
| | 35. Salty fish (cod, dried charales) | 1 ration (90 g) | |
| | 36. Canned fish (tuna, sardine) or shellfish in water | ½ can (55g) | |
| | 37. Canned fish (tuna, sardine) or shellfish in oil | ½ can (55g) | |
| | 38. Shellfish (shrimp, prawn) | 10 piece (68 g) | |
| | 38.1 River prawn | 10 piece (68 g) | |
| | 39. Octopus or squid | 1 ration (100 g) | |
| | 40. Oysters, clams, mussels | 4 pieces (58 g) | |
| | 40.1 Insects (maguey worms, crickets) | 1 portion (35 g) | |
| | 41. Frozen vegetables | ½ cup (46 g) | |
| | 42. Spinach, chard or purslane | 1/2 cup (30 g) | |
| | 43. Broccoli or cauliflower | ½ cup (108 g) | |
| | 44. Lettuce, cabbage, cabbage or kale | ½ cup (25 g) | |
| | 45. Red tomato raw or in sauce | 1 piece (60 g) | |
| | 46. Carrot | ½ piece (64g) | |
| | 47. Zucchini | 1 piece (91 g) | |
| | 48. Pumpkin | ½ cup (110 g) | |
| | 49. Green beans or peas | ½ cup (63 g) | |
| les | 50. Cucumber | 1 piece (104 g) | |
| Vegetables | 51. Celery | ½ cup (45 g) | |
| ge | 52. Beetroot | ½ piece (39 g) | |
| > | 53. Eggplant | ½ cup (50 g) | |
| | 54. Asparagus | 3 piece (45 g) | |
| | 55. Onion | ½ cup (29 g) | |
| | 56. Green tomato, raw or in sauce | 4 pieces (69 g) | |
| | 57. Mushrooms | ½ cup (70 g) | |
| | 57.1 Huitlacoche | 1/3 cup (66 g) | |
| | 58. Chayote | ½ cup (80 g) | |
| | 59. Jicama | ½ cup (60 g) | |
| | 60. Cooked, raw or roasted nopales (cactus) | ½ cup (75g) | |
| | 61. Bell pepper | 1/2 piece (32 g) | |

| | 62. Poblano Chile | 1/2 piece (32 g) |
|---|---|---|
| | 62.1 Quelites | ½ cup (66 g) |
| | 62.2 Purslane | 1 cup (115 g) |
| | 63. Hot peppers (jalapeño, serrano, habanero) | 1 piece (30 g) |
| | 64. Garlic | ½ piece (1 g) |
| | 65. Coriander, parsley, oregano, basil, bay leaf | 1 pinch (6 g) |
| | 66. Orange (not in juice) | 1 piece (76 g) |
| | 67. Grapefruit (not in juice) | 1 piece (76 g) |
| | 68. Tangerines (not in juice) | 1 piece (76 g) |
| | 69. Lemon | 1 piece (38 g) |
| | 70. Lime (not in juice) | 1 piece (49 g) |
| | 71. Banana (not fried) | 1 piece (49 g) 1 piece (108 g) |
| | 72. Apple | 1 piece (106 g) |
| | 73. Pear | 1 piece (160 g) 1 piece (162 g) |
| | 74. Strawberries | 6 pieces (68 g) |
| | 75. Blueberry | ½ cup (49 g) |
| | 76. Raspberry | ½ cup (61 g) |
| | 77. Blackberry | ½ cup (72 g) |
| | 78. Creole plum | 2 pieces (105 g) |
| | 78.1 Capulín | 2 pieces (103 g) 1 cup (32 g) |
| | 78.1 Capulin 78.2 Nance | 5 pieces (15 g) |
| Fruits | 79. Cherries | 4 pieces (18 g) |
| Ξ | | |
| | 80. Peach | 1 piece (77 g) |
| | 81. Nectarine | 1 piece (124 g) |
| | 82. Watermelon | 1 cup (160 g) |
| | 83. Cantaloupe | 1 cup (160 g) |
| | 84. Papaya | 1 cup (140 g) |
| | 85. Kiwi | 1 piece (76 g) |
| | 86. Grapes | 18 pieces (86 g) |
| | 87. Mango | ½ piece (110 g) |
| | 88. Guava | 2 pieces (83 g) |
| | 89. Tuna | 1 piece (70 g) |
| | 90. Pitaya | 1 piece (50 g) |
| | 91. Guanabana | ½ piece (175 g) |
| | 92. Pineapple | 1 cup (165 g) |
| | 93. Canned fruit in syrup | ½ cup (124 g) |
| | 94. Dehydrated fruit (blueberries, raisins, dates, prune) | 10 pieces (20 g) |
| | 95. Almonds | 10 pieces (12 g) |
| si | 96. Raw peanuts | 14 pieces (12 g) |
| Protein oils | 96.1 Peanuts (Japanese, enchiladas, with salt) | 14 pieces (12 g) |
| tein | 97. Nuts | 7 halvez (10 g) |
| 2ro | 98. Pistachios, hazelnuts, pine nuts | 18 pieces (13 g) |
| Ι " | 98.1 Dried beans | 18 pieces (13 g) |
| | 99. Sunflower or hemp seeds | 1 tablespoon (10 g) |

| | 99.1 Pumpkin seeds | 1 tablespoon (10 g) |
|---|---|---|
| | 100. Chia seeds | 1 teaspoon (3 g) |
| | 100.1 Flax | 1 teaspoon (3 g) |
| | 101. Peanut or almond butter | 1 tablespoon (15 g) |
| | 102. Cooked beans | ½ cup (99 g) |
| | 103. Refried beans | ½ cup (99 g) |
| es | 104. Cooked lentils | ½ cup (99 g) |
| Legumes | 105. Cooked chickpeas | ½ cup (82 g) |
| eg , | 105.1 Baked beans | ½ cup (99 g) |
| | 106. Chickpea hummus | 4 tablespoon (60 g) |
| | 107. Textured soy | 1/2 cup (30 g) |
| | 108. Corn tortilla | 1 piece (30 g) |
| | 10.8.1 Corn dough | 1 ball (45 g) |
| | 109. Corn | 1 piece (116 g) |
| | 110. Baked or boiled potato | 1 piece (136 g) |
| | 111. Flour tortilla | 1 piece (28 g) |
| | 112. Wholemeal flour tortilla | 1 piece (28 g) |
| | 113. Bolillo, birote or telera (not in cake) | ½ piece (30 g) |
| | 114. White bread or toast white bread (apart from sandwich) | 1 slice (27 g) |
| | 115. Whole wheat bread or toast whole wheat bread (apart from | 1 slice (25 g) |
| | sandwich) | |
| | 116. Unsweetened box cereal | 1 cup (25 g) |
| | 117. Sweetened box cereal | 1 cup (25 g) |
| eal | 118. Whole wheat box cereal | 1 cup (25 g) |
| cer | 119. Pasta (noodles, macaroni, spaghetti) | ½ cup (60 g) |
| Fat-free cereal | 120. Oatmeal (flaked, cooked in water) | ½ cup (20 g) |
| t-fr | 121. Cooked oatmeal with milk and sugar (drink or solid) | 1 cup (240 ml) |
| Fa | 122. Cooked white rice or Mexican cooked white rice | ½ cup (94 g) |
| | 123. Brown or wild rice | ½ cup (94 g) |
| | 124. Natural puffed rice or puffed rice cake | ½ cup (17 g) |
| | 125. Unsweetened amaranth | ½ cup (32 g) |
| | 125.1 Sweetened amaranth or amaranth bar | ½ cup (32 g) |
| | 126. Cooked sweet potato | ½ cup (103 g) |
| | 127. Sweet potato cooked with sugar | ½ cup (103 g) |
| | 128. Quinoa | ½ cup (40 g) |
| | 129. Marías or animals shape biscuits | 5 pieces (19 g) |
| | 130. Whole meal or fibre biscuits (sweet or salty type) | 1 sweet or 9 salty (45<br>g) |
| | 131. Salty biscuits | 4 pieces (16 g) |
| | 132. Baked Maize toast | 1 piece (10 g) |
| | 133. Fried Maize toast | 1 piece (12 g) |
| y | 134. Packaged sweet biscuits | 2 piece (21 g) |
| Fatty<br>cereal | 135. Granola bar | 1 piece (35g) |
| E 2 | 136. Granola with nuts | 3 tablespoons (21 g) |

| | 137. Hot cake or waffle | 1 piece (50 g) | T I | | |
|---|---|---|---|---|---|
| | 138. Industrialized bread (donuts, shortcakes) | 1 piece (30 g) | | | |
| | 139. Industrialized bread with chocolate | 1 piece (50 g) | | | |
| | 140. Sweet bread (conchas, orejas, polvorón) | 1 piece (63 g) | | | |
| | 141. Cake or pay (thick slice) | 1 slice (56 g) | | | |
| | 142. Homemade breads or rosca de reyes | 1 slice (56 g) | | | |
| | 143. Packaged chips | 1 bag (55 g) | | | |
| | 144. Packaged Maize snack | 1 bag (58 g) | | | |
| | 145. French fries or home fries | 4 pieces (20 g) | | | |
| | 146. Wheat churritos | 1 bag (50 g) | | | |
| | 147. Popcorn (homemade, microwave, cinema) | ½ bag (40 g) | | | $\overline{}$ |
| | 148. Oil spray | 5 sprays (5 g) | | | |
| | 149. Olive oil | 1 teaspoonful (5 g) | | | |
| | 150. Avocado oil | 1 teaspoonful (5 g) | | | |
| | 151. Maize oil | 1 teaspoonful (5 g) | | | |
| | 152. Coconut oil | 1 teaspoonful (5 g) | | | |
| | 153. Sunflower oil | 1 teaspoonful (5 g) | | | |
| | 154. Soy oil | 1 teaspoonful (5 g) | | | |
| ×. | 155. Canola oil | 1 teaspoonful (5 g) | | | |
| Protein oils | 156. Safflower oil | 1 teaspoonful (5 g) | | | |
| ein | 157. Olives | 8 pieces (24 g) | | | |
| rot | 158. Chopped coconut | 1 strip (16 g) | | | |
| Ъ | 159. Avocado or guacamole | ½ pieces (46 g) | | | |
| | 160. Mayonnaise, dressing or vinaigrette | 1 teaspoonful (5 g) | | | |
| | 161. Margarine | 1 teaspoonful (5 g) | | | |
| | 162. Butter | 1 teaspoonful (5 g) | | | |
| | 163. Lard | 1 teaspoonful (5 g) | | | |
| | 164. Vegetable shortening | 1 teaspoonful (5 g) | | | |
| | 165. Cream cheese | 1 tablespoon (15 g) | | - | |
| | 166. Cream, nata or jocoque | 1 tablespoon (15 g) | | | |
| | 167. Sugar | 1 teaspoonful (4 g) | | | |
| | 168. Honey | 1 teaspoonful (7 g) | | | |
| fat | 169. Maple syrup | 1 teaspoonful (7 g) | | $\rightarrow$ | |
| Ħ | 170. Cajeta | 1 tablespoon (15 g) | | | |
| tho | 171. Hazelnut cream | 1 tablespoon (15 g) | | | |
| W. | 172. Condensed milk | 1 tablespoon (15 g) | | | |
| pu | 173. Piloncillo (brown sugar) | 1 portion (10 g) | | - | |
| E a | 174. Jams | 1 tablespoon (17 g) | | | |
| Sugars with and without fat | 175. Packaged candy (i.e. popsicles, solid sweets, jelly beans) | 1 - 5 pieces (20 g) | | | |
| ars | 176. Chocolates | 1 bar (15 g) | | | |
| ı g | 177. Cocoa powder for chocolate milk | 1 tablespoon (15 g) | | | |
| SO . | 178. Ice cream or ice cream popsicle | 1 scoop/piece (96 g) | | | |
| | 179. Water-based ice cream or ice cold water palette | 1 scoop/piece (65 g) | | | |
| | 180. Tapioca (cooked in caramel or milk) | ½ cup (147 g) | | | |

| | 181. Gelatin in water or milk | 1 piece (125 ml) | 1 | |
|---|---|---|---|---|
| | 182. Mexican candy ( <i>Ate, cocada, marzipan, palanqueta</i> | 1 piece (28 g) | | |
| | (peanut or walnut), milk candy) | 1 piece (28 g) | | |
| | 183. Fried or honeyed bananas | 1 piece (123.5 g) | | |
| | 184. Pizza | 1 slice (100 g) | | |
| | 185. Burger | 1 piece (235 g) | | |
| | 186. Hot dog | 1 piece (156 g) | | |
| Fast food | 187. Ham sandwich | 1 piece (128 g) | | |
| t fo | 188. Instant soup | 1 piece (64 g) | | |
| Fas | 189. Sushi | 4 rolls (75 g) | | |
| | 190. Chicken wings | 1 piece (51 g) | | |
| | 191. Baguette or panini | 1 piece (208 g) | | |
| | 192. Envelope soups and creams | 1 plate (100 g) | | |
| | 193. Chilaquiles with beef | 1 cup (160 g) | | |
| | 193. Chilaquiles with egg and/or chicken but without beef | 1 cup (160 g) | | |
| | 193.1 Mexican style egg (tomato, onion, chili, nopal) | 1 plate (220 g) | | |
| | 194. Offal | 1 plate (300 g) | | |
| | 195. Corn tortilla quesadillas without meats | 1 piece (60 g) | | |
| | 195.1 Corn tortilla quesadillas with meats | 1 piece (60 g) | | |
| | 196. Flour tortilla quesadillas | 1 piece (60 g) | | |
| | 197. Torta (marinated, meat, drowned) | 1 piece (197 g) | | |
| | 197.1 Panela cake or beans (not meat) | 1 piece (197 g) | | |
| | 198. Meat tamale (beef, pork, chicken) | 1 piece (200 g) | | |
| | 198.1 Chicken tamale | 1 piece (200 g) | | |
| | 198.2 Cheese tamale | 1 piece (200 g) | | |
| | 198.3 Tamale of rajas or ash (beans) | 1 piece (200 g) | | |
| Mexican food | 199. Sweet tamale (corn, fruits) | 1 piece (172 g) | | |
| l g | 200. Mole with chicken | 1 plate (334 g) | | $\perp$ |
| [ <u>s</u> | 201. Pork pozole | 1 plate (300 g) | | |
| [ex] | 201.1 Chicken pozole | 1 plate (300 g) | | _ |
| ≥ | 201.2 Vegetarian pozole (mushrooms) | 1 plate (300 g) | | |
| | 202. Sopitos with beef or pork | 1 piece (75 g) | | |
| | 202.1 Sopitos of beans or chicken (no red meat) | 1 piece (75 g) | | |
| | 202.1 Enchiladas with beef or pork | 1 piece (75 g) | | |
| | 202.2 Chicken or cheese enchilada (no red meat) | 1 piece (75 g) | | |
| | 202.2 Flautas with beef or pork | 1 piece (75 g) | | |
| | 202.3 Chicken or cheese flautas (no red meat) | 1 piece (75 g) | | |
| | 203. Natural vegetable soups, broths or creams | 1 plate (393 g) | | |
| | 204. Beef tacos | 1 piece (75 g) | | |
| | 204.1 Pork tacos (adobado, al pastor) | 1 piece (75 g) | | |
| | 204.2 Beans taco | 1 piece (60 g) | | |
| | 204.3 Chicken or fish tacos | 1 piece (75 g) | | |
| | 205. Beef burrito | 1 piece (100 g) | | |
| | 205.1 Meatless Bean Burrito | 1 piece (100 g) | | |

| 1 1 1 1 20.5 Tosts with beaus or chicken 1 1 1 20.5 1 20.5 1 20.5 20.5 | | 205.2 Toast with beef or pork | 1 large toast (174g) |
|---|---|---|---|
| 200. Rice pending | | | |
| 207. Flans, pricellale, postand | | | |
| 208. Captrostada | | | |
| 209. Staffed or sugared churros | | | |
| 210. Corn atole in water | | | |
| 211. Corn atole in milk or champurado 1 cup (240 ml) | | | |
| 212. Ketchup or eanned tomato puree | | 211. Corn atole in milk or champurrado | |
| 213. Bottled hot sauce | | • | |
| 11 suspoonful (5 g) 1 pinch (2 g) 215. Salt 1 pinch (2 g) 215. Salt 1 pinch (2 g) 216. Say sance 1 reaspoonful (5 mi) 217. Vanilla, pepper, cinnamon, ginger, turmeric, curry, cloves, enise 1 reaspoonful (5 g) 218. Coffee creamer 1 feaspoonful (5 g) 229. Soft drink or drink with sugar 1 feaspoonful (5 g) 229. Soft drink or drink without sugar 1 feaspoonful (5 g) 229. Soft drink or drink without sugar 1 cup (240 mi) 221. Fresh fruit water without sugar 1 cup (240 mi) 222. Natural furit piuce (corange, grapefruit) 1 cup (240 mi) 223. Industrialized fruit piuce 1 feaspoonful (5 g) 224. Sports drink (Gatorade, etc) 1 bottle (690 mi) 225. Tejuino 2 cups (418 mi) 225. Tejuino 2 cups (418 mi) 225. Tituba 1 cup (240 mi) 225. Cappaceinos or lates 1 cup (240 mi) 227. Coffee pot 1 cup (240 mi) 228. Cappaceinos or lates 1 cup (240 mi) 229. Frappuccinos or milk shakes 2 cups (480 mi) 229. Frappuccinos or milk shakes 2 cups (480 mi) 229. Tejuinamon 1 cup (240 mi) 229. Tejuinamon 229. Tejuinamon 229. Tejuinamon 229. Tejui | | | |
| anise 1 teaspoonful (5 g) | nts | 214. Mustard | |
| anise 1 teaspoonful (5 g) | me | 215. Salt | |
| anise 218. Coffee creamer 1 teaspoonful (5 g) | je j | 216. Soy sauce | |
| anise 218. Coffee creamer 1 teaspoonful (5 g) | J | • | |
| 219. Soft drink or drink with sugar 1 bottle (600 ml) 220. Soft drink or drink without sugar or light 1 bottle (600 ml) 221. Fresh fruit water with sugar 1 cup (240 ml) 221. Fresh fruit water without sugar 1 cup (240 ml) 222. Natural fruit juice (orange, grapefruit) 1 cup (240 ml) 223. Industrialized fruit juice 1 bottle (240 ml) 225. Tejuino 2 cups (418 ml) 225. Tejuino 2 cups (418 ml) 225. Tejuino 2 cups (418 ml) 226. Soluble or American coffee 1 cup (240 ml) 227. Coffee pot 1 cup (240 ml) 228. Cappuccinos or lattes 1 cup (240 ml) 229. Frappuccinos or lattes 1 cup (240 ml) 229. Frappuccinos or lattes 1 cup (240 ml) 229. Frappuccinos or lattes 1 cup (240 ml) 229. Frappuccinos or milk shakes 2 cups (480 ml) 229. Frappuccinos or milk shakes 1 cup (240 ml) 229. Frappuccinos or milk shakes 1 cup (240 ml) 229. Frappuccinos or milk shakes 1 cup (240 ml) 229. Frappuccinos or milk shakes 1 cup (240 ml) 229. Frappuccinos or milk shakes 2 cups (480 ml) 220. Chocolate in water 1 cup (240 ml) 220. Tea or cinnamon 1 cup (240 ml) | | anise | |
| 220. Soft drink or drink without sugar or light 1 bottle (600 ml) 221. Fresh fruit water with sugar 1 cup (240 ml) 221. I Fresh fruit water without sugar 1 cup (240 ml) 222. Natural fruit juice (orange, grapefruit) 1 cup (240 ml) 223. Industrialized fruit juice 1 bottle (240 ml) 224. Sports drink (Gatorade, etc) 1 bottle (600 ml) 225. Tejuino 2 cups (418 ml) 225. Tejuino 2 cups (418 ml) 225. Tejuino 2 cups (418 ml) 225. Zaspados 2 cups (418 ml) 225. Zaspados 2 cups (418 ml) 227. Coffee pot 1 cup (240 ml) 228. Cappucinos or lattes 1 cup (240 ml) 229. Frappuccinos or milk shakes 2 cups (480 ml) 229. Frappuccinos or milk shakes 2 cups (480 ml) 230. Chocolate in water 1 cup (240 ml) 231. Milk chocolate 1 cup (240 ml) 232. Tea or cinnamon 1 cup (240 ml) 233. Natural water 1 cup (240 ml) 234. Red wine 1 glass (100 ml) 234. Red wine 1 glass (100 ml) 234. Red wine 1 glass (100 ml) 234. Red wine 1 glass (100 ml) 234. Red wine 1 glass (100 ml) 235. Red wine 1 glass (100 ml) 235. Red wine 1 glass (100 ml) 236. Red wine 1 glass (100 ml) 236. Red wine 1 glass (100 ml) 236. Red wine 1 glass (100 ml) 237. Red wine 1 glass (100 ml) 238. Red wine 1 glass (100 ml) 239. Red wine 1 gl | | | |
| 221. Fresh fruit water without sugar 1 cup (240 ml) | | <u> </u> | |
| 221.1 Fresh fruit water without sugar 1 cup (240 ml) 222. Natural fruit juice (orange, grapefruit) 1 cup (240 ml) 223. Industrialized fruit juice 1 bottle (600 ml) 224. Sports drink (Gatorade, etc) 1 bottle (600 ml) 225. Tejuino 2 cups (418 ml) 225.1 Tuba 1 cup (240 ml) 225.2 Raspados 2 cups (418 ml) 226. Soluble or American coffee 1 cup (240 ml) 227. Coffee pot 1 cup (240 ml) 228. Cappuccinos or lattes 1 cup (240 ml) 229. Frappuccinos or milk shakes 2 cups (480 ml) 229. Frappuccinos or milk shakes 2 cups (480 ml) 220. Chocolate in water 1 cup (240 ml) 221. Milk chocolate 1 cup (240 ml) 222. Tea or cinnamon 1 cup (240 ml) 223. Natural water 1 cup (240 ml) 223. Natural water 1 cup (240 ml) 223. Natural water 1 cup (240 ml) 223. Natural water 1 cup (240 ml) 224. Red wine 1 glass (100 ml) 224. Red wine 1 glass (100 ml) 225. Tea or cinnamon 1 cup (240 ml) 225. Tea or cinnamon 225. Tea or | | | |
| 222. Natural fruit juice (orange, grapefruit) 223. Industrialized fruit juice 1 bottle (240 ml) 224. Sports drink (Gatorade, etc) 1 bottle (660 ml) 225. Tejuino 226. Soluble or American coffee 1 cup (240 ml) 225. Raspados 2 cups (418 ml) 225. Raspados 2 cups (418 ml) 226. Soluble or American coffee 1 cup (240 ml) 227. Coffee pot 228. Cappuccinos or lattes 1 cup (240 ml) 229. Frappuccinos or milk shakes 2 cups (480 ml) 230. Chocolate in water 1 cup (240 ml) 231. Milk chocolate 1 cup (240 ml) 232. Tea or cinnamon 1 cup (240 ml) 233. Natural water 1 cup (240 ml) 234. Red wine 1 glass (100 ml) | | | |
| 223. Industrialized fruit juice 1 bottle (240 ml) | | <u> </u> | |
| 224. Sports drink (Gatorade, etc) 1 bottle (600 ml) 2 cups (418 ml) 2 cups (418 ml) 1 cup (240 ml) 225. I Raspados 2 cups (418 ml) 226. Soluble or American coffee 1 cup (240 ml) 227. Coffee pot 1 cup (240 ml) 228. Cappuccinos or lattes 1 cup (240 ml) 229. Frappuccinos or milk shakes 2 cups (480 ml) 230. Chocolate in water 1 cup (240 ml) 231. Milk chocolate 1 cup (240 ml) 232. Tea or cinnamon 1 cup (240 ml) 233. Natural water 1 cup (240 ml) 234. Red wine 1 glass (100 ml) | | 3 ( 0.0 1 ) | |
| 225. Tejuino 2 cups (418 ml) 225.1 Tuba 1 cup (240 ml) 225.2 Raspados 2 cups (418 ml) 226. Soluble or American coffee 1 cup (240 ml) 227. Coffee pot 1 cup (240 ml) 228. Cappuccinos or lattes 1 cup (240 ml) 229. Frappuccinos or milk shakes 2 cups (480 ml) 229. Frappuccinos or milk shakes 1 cup (240 ml) 231. Milk chocolate 1 cup (240 ml) 232. Tea or cinnamon 1 cup (240 ml) 233. Natural water 1 cup (240 ml) 234. Red wine 1 glass (100 ml) | | 2 | |
| Composition | | | |
| 227. Coffee pot 1 cup (240 ml) 228. Cappuccinos or lattes 1 cup (240 ml) 229. Frappuccinos or milk shakes 2 cups (480 ml) 230. Chocolate in water 1 cup (240 ml) 231. Milk chocolate 1 cup (240 ml) 232. Tea or cinnamon 1 cup (240 ml) 233. Natural water 1 cup (240 ml) 234. Red wine 1 glass (100 ml) | ses | | |
| 227. Coffee pot 1 cup (240 ml) 228. Cappuccinos or lattes 1 cup (240 ml) 229. Frappuccinos or milk shakes 2 cups (480 ml) 230. Chocolate in water 1 cup (240 ml) 231. Milk chocolate 1 cup (240 ml) 232. Tea or cinnamon 1 cup (240 ml) 233. Natural water 1 cup (240 ml) 234. Red wine 1 glass (100 ml) | rag | | |
| 227. Coffee pot 1 cup (240 ml) 228. Cappuccinos or lattes 1 cup (240 ml) 229. Frappuccinos or milk shakes 2 cups (480 ml) 230. Chocolate in water 1 cup (240 ml) 231. Milk chocolate 1 cup (240 ml) 232. Tea or cinnamon 1 cup (240 ml) 233. Natural water 1 cup (240 ml) 234. Red wine 1 glass (100 ml) | eve | • | |
| 228. Cappuccinos or lattes 1 cup (240 ml) 229. Frappuccinos or milk shakes 2 cups (480 ml) 230. Chocolate in water 1 cup (240 ml) 231. Milk chocolate 1 cup (240 ml) 232. Tea or cinnamon 1 cup (240 ml) 233. Natural water 1 cup (240 ml) 234. Red wine 1 glass (100 ml) | ğ | | |
| 229. Frappuccinos or milk shakes 2 cups (480 ml) 230. Chocolate in water 1 cup (240 ml) 231. Milk chocolate 1 cup (240 ml) 232. Tea or cinnamon 1 cup (240 ml) 233. Natural water 1 cup (240 ml) 234. Red wine 1 glass (100 ml) | | - | |
| 230. Chocolate in water 1 cup (240 ml) | | | |
| 231. Milk chocolate | | • • | |
| 232. Tea or cinnamon 1 cup (240 ml) | | | |
| 233. Natural water 1 cup (240 ml) 234. Red wine 1 glass (100 ml) | | | |
| 234. Red wine 1 glass (100 ml) | | | |
| 235. White or rosé wine 1 glass (100 ml) 236. Beer 1 can or bottle (356 ml) 237. Spirits: whiskey, vodka, gin, cognac, tequila, mezcal, rum, 1 shot (60 ml) | | | |
| 236. Beer 1 can or bottle (356 ml) 237. Spirits: whiskey, vodka, gin, cognac, tequila, mezcal, rum, 1 shot (60 ml) | sk | | |
| 237. Spirits: whiskey, vodka, gin, cognac, tequila, mezcal, rum, 1 shot (60 ml) | i <u>f</u> | | 1 can or bottle (356 ml) |
| • brandy | olic | 237. Spirits: whiskey, vodka, gin, cognac, tequila, mezcal, rum, brandy | 1 shot (60 ml) |
| 238. Punch (pomegranate, raspberry) 1 glass (80 ml) | e de la companya de l | 238. Punch (pomegranate, raspberry) | 1 glass (80 ml) |
| 239. Rompope 1 glass (80 ml) | Ā | 239. Rompope | 1 glass (80 ml) |
| 240. Pulque, tepache or honey water 1 glass (80 ml) | | 240. Pulque, tepache or honey water | 1 glass (80 ml) |
| 241. Protein supplement 1 scoop (40 g) | _ q | 241. Protein supplement | 1 scoop (40 g) |
| 242. Estevia 1 sachet (3g) | _ <del>_</del> = | 242. Estevia | 1 sachet (3g) |

| | 243. Splenda® or Canderel® | 1 sachet (3g) |
|---|---|---|
| | 244. Multivitamin supplements (place mark) | 1 capsule |
| | 245. Kéfir | 1 cup (240 ml) |
| ge | 246. Kombucha (Fermented tea) | 1 cup (240 ml) |
| Ę. | 247. Tempeh (Fermented soy) | 1 cup (240 ml) |
| eq | 248. Natto (Fermented soy) | 1 cup (240 ml) |
| ent | 249. Miso (Fermented soybean paste) | 1 cup (240 ml) |
| E | 250. Kimchi (Fermented vegetables) | 1 cup (240 ml) |
| Fe | 251. Sourdough bread (Sourdough bread) | 1 cup (240 ml) |
| | 252. Saurkraut (Fermented cabbage) | 1 cup (240 ml) |

Note: foods colored blue corresponds to those that will be included in the intervention program and correspond to those presented in Table A6.5, where the frequency and quantity of consumption to be promoted are specified. FCFQ adapted from: Lares-Michel, M.; Housni, F. E.; Aguilera Cervantes, V. G.; Michel Nava, R. M. Nutriecology: A Mexican web-based nutritional ecologic software for the assessment of diet, dietary pattern, diet quality, and dietary environmental impact. Nutrients (under revision).

Supplementary Material 4. COM-B questionnaire including nutritional-sustainable knowledge questions

This questionnaire will be modified based on the issues addressed during the development of the program, as well as based on the execution of the pilot test, where multiple options will be established for data analysis. However, the format to be used and the questions determined so far are presented below, which incorporate the elements of the COM-B model, which include capacity, opportunity, and motivation (14). Likewise, questions on sustainable food consumption were integrated, according to the questionnaire by Verain et al. (62).

Table SM4.1. COM-B questionnaire including nutritional-sustainable knowledge questions

| COM-B questionnaire | | | |
|---|---|---|---|
| Participant number: | | | |
| Date: | | | |
| COM-B dimension | Answer | Mark your answer | Explain your answer |
| Capability | | | |
| Knowledge of general nutrition and susta | inability | | |
| | Yes | | |
| Do you know which food groups exist? | No | | |
| | | write them down please. | |
| | Yes | | |
| Do you know what foods contain carbohydrates? | No | | |
| | | write them down please. | |
| | Yes | | |
| Do you know what foods contain fat? | No | | |
| | | write them down please. | |
| | Yes | | |
| Do you know what foods contain protein? | No | | |
| | | write them down please. | |
| | Yes | | |
| Did you know that the food you eat requires high amounts of water during its production? | No | | |
| | | your answer please | |
| Did you know that the food you eat generates greenhouse gas emissions during its production, which promote | Yes | | |
| climate change? | No | | |

| | Explain your answer please |
|---|---|
| W (C. 1.1. d.) | Yes |
| What foods do you think use more water during their production? | No |
| | If you know, write them down please. |
| | Yes |
| What foods do you think generate more greenhouse gas emissions during their production? | No |
| | If you know, write them down please. |
| | Yes |
| Do you consider that the traditional Mexican diet is healthy? | No |
| | Explain your answer please |
| | Yes |
| Do you consider that the tortilla is "fattening"? | No |
| , | Explain your answer please |
| | Yes |
| Do you consider that buying food in local markets or markets is frowned upon? | No |
| Do you consider that caying root in rotal markets of markets is nowned upon. | Explain your answer please |
| | Yes |
| Do you consider it a better entire to buy your food in our employed then in local markets? | No |
| Do you consider it a better option to buy your food in supermarkets than in local markets? | <u> </u> |
| | Explain your answer please |
| | Yes |
| If you knew all the environmental impacts of your diet, would you change it? | No |
| | Explain your answer please |
| | Yes |
| Would you be willing to eat less red meat if you knew that it had a high environmental impact? | No |
| | Explain your answer please |
| | Yes |
| Do you know what sustainable diets are? | No |
| | Explain your answer please |
| Specific nutrition and sustainability knowledge | |
| Aspect | Write your answer please |
| Please mention the benefits of physical activity | |
| Mention what is the recommended amount of physical activity to perform per day | |
| Please mention the benefits of consuming a traditional Mexican diet | |
| Mention what is the recommended amount to consume of portions of Mexican food per day | |
| Please mention the benefits of consuming fruits and vegetables | |
| Mention what is the recommended amount to consume of servings of fruits and vegetables per day | |
| Please mention the benefits of consuming whole grains | |
| Mention what is the recommended amount to consume of servings of whole grains per day | |
| Please mention the benefits of consuming legumes | <u> </u> |
| Mention what is the recommended amount to consume portions of legumes per day | |
| Please mention the benefits of consuming seeds and healthy fats | |
| Mention what is the recommended amount to consume of portions of seeds and healthy fats per day | |
| Please mention the benefits of consuming dairy in adequate amounts | |
| Mention what is the recommended amount to consume of dairy portions per day | |

| Please mention the benefits of consuming eggs in adequate amounts Mention what is the recommended amount to consume of servings of eggs per day Please mention the benefits of consuming fish and shellfish in adequate amounts Mention what is the recommended amount to consume of portions of fish and shellfish per day Please mention the benefits of consuming chicken in adequate amounts Mention what is the recommended amount to consume chicken portions per day Please mention the benefits of avoiding red and processed meats Mention what is the recommended amount to consume of portions of red and processed meats Please mention the benefits of avoiding ultra-processed foods Mention what is the recommended amount to consume of portions of ultra-processed foods per day Please mention the benefits of avoiding added sugar, foods high in trans and saturated fats Mention what is the recommended amount to consume of portions of ultra-processed foods per day Please mention the benefits of avoiding added sugar, foods high in trans and saturated fats Mention what is the recommended amount to consume of portions of added sugar, foods high in trans and saturated fats Food preparation skills Do you know how to cook? Yes / No Does it have a kitchen equipped with a stove? Yes / No Does it have a kitchen equipped with a refrigerator? Yes / No |
|---|
| Please mention the benefits of consuming fish and shellfish in adequate amounts Mention what is the recommended amount to consume of portions of fish and shellfish per day Please mention the benefits of consuming chicken in adequate amounts Mention what is the recommended amount to consume chicken portions per day Please mention the benefits of avoiding red and processed meats Mention what is the recommended amount to consume of portions of red and processed meats Please mention the benefits of avoiding ultra-processed foods Mention what is the recommended amount to consume of portions of ultra-processed foods per day Please mention the benefits of avoiding added sugar, foods high in trans and saturated fats Mention what is the recommended amount to consume of portions of added sugar, foods high in trans and saturated fats Mention what is the recommended amount to consume of portions of added sugar, foods high in trans and saturated fats Food preparation skills Do you know how to cook? Yes / No Preparation capacity Does it have a kitchen equipped with a stove? Yes / No |
| Mention what is the recommended amount to consume of portions of fish and shellfish per day Please mention the benefits of consuming chicken in adequate amounts Mention what is the recommended amount to consume chicken portions per day Please mention the benefits of avoiding red and processed meats Mention what is the recommended amount to consume of portions of red and processed meats Please mention the benefits of avoiding ultra-processed foods Mention what is the recommended amount to consume of portions of ultra-processed foods per day Please mention the benefits of avoiding added sugar, foods high in trans and saturated fats Mention what is the recommended amount to consume of portions of added sugar, foods high in trans and saturated fats Food preparation skills To bo you know how to cook? If the answer was yes, what foods do you know how to cook? Preparation capacity Does it have a kitchen equipped with a stove? Yes / No |
| Please mention the benefits of consuming chicken in adequate amounts Mention what is the recommended amount to consume chicken portions per day Please mention the benefits of avoiding red and processed meats Mention what is the recommended amount to consume of portions of red and processed meats Please mention the benefits of avoiding ultra-processed foods Mention what is the recommended amount to consume of portions of ultra-processed foods per day Please mention the benefits of avoiding added sugar, foods high in trans and saturated fats Mention what is the recommended amount to consume of portions of added sugar, foods high in trans and saturated fats Food preparation skills Do you know how to cook? Yes / No Preparation capacity Does it have a kitchen equipped with a stove? Yes / No |
| Mention what is the recommended amount to consume chicken portions per day Please mention the benefits of avoiding red and processed meats Mention what is the recommended amount to consume of portions of red and processed meats Please mention the benefits of avoiding ultra-processed foods Mention what is the recommended amount to consume of portions of ultra-processed foods per day Please mention the benefits of avoiding added sugar, foods high in trans and saturated fats Mention what is the recommended amount to consume of portions of added sugar, foods high in trans and saturated fats Food preparation skills Do you know how to cook? Yes / No Preparation capacity Does it have a kitchen equipped with a stove? Yes / No |
| Please mention the benefits of avoiding red and processed meats Mention what is the recommended amount to consume of portions of red and processed meats Please mention the benefits of avoiding ultra-processed foods Mention what is the recommended amount to consume of portions of ultra-processed foods per day Please mention the benefits of avoiding added sugar, foods high in trans and saturated fats Mention what is the recommended amount to consume of portions of added sugar, foods high in trans and saturated fats Food preparation skills Do you know how to cook? Yes / No If the answer was yes, what foods do you know how to cook? Preparation capacity Does it have a kitchen equipped with a stove? Yes / No |
| Mention what is the recommended amount to consume of portions of red and processed meats Please mention the benefits of avoiding ultra-processed foods Mention what is the recommended amount to consume of portions of ultra-processed foods per day Please mention the benefits of avoiding added sugar, foods high in trans and saturated fats Mention what is the recommended amount to consume of portions of added sugar, foods high in trans and saturated fats Food preparation skills Do you know how to cook? Yes / No If the answer was yes, what foods do you know how to cook? Preparation capacity Does it have a kitchen equipped with a stove? Yes / No |
| Please mention the benefits of avoiding ultra-processed foods Mention what is the recommended amount to consume of portions of ultra-processed foods per day Please mention the benefits of avoiding added sugar, foods high in trans and saturated fats Mention what is the recommended amount to consume of portions of added sugar, foods high in trans and saturated fats Food preparation skills Do you know how to cook? Yes / No If the answer was yes, what foods do you know how to cook? Preparation capacity Does it have a kitchen equipped with a stove? Yes / No |
| Mention what is the recommended amount to consume of portions of ultra-processed foods per day Please mention the benefits of avoiding added sugar, foods high in trans and saturated fats Mention what is the recommended amount to consume of portions of added sugar, foods high in trans and saturated fats Food preparation skills Do you know how to cook? Yes / No If the answer was yes, what foods do you know how to cook? Preparation capacity Does it have a kitchen equipped with a stove? Yes / No |
| Please mention the benefits of avoiding added sugar, foods high in trans and saturated fats Mention what is the recommended amount to consume of portions of added sugar, foods high in trans and saturated fats Food preparation skills Do you know how to cook? Yes / No If the answer was yes, what foods do you know how to cook? Preparation capacity Does it have a kitchen equipped with a stove? Yes / No |
| Mention what is the recommended amount to consume of portions of added sugar, foods high in trans and saturated fats Food preparation skills Do you know how to cook? Yes / No If the answer was yes, what foods do you know how to cook? Preparation capacity Does it have a kitchen equipped with a stove? Yes / No |
| Food preparation skills Do you know how to cook? Yes / No If the answer was yes, what foods do you know how to cook? Preparation capacity Does it have a kitchen equipped with a stove? Yes / No |
| Food preparation skills Do you know how to cook? If the answer was yes, what foods do you know how to cook? Preparation capacity Does it have a kitchen equipped with a stove? Yes / No |
| Do you know how to cook? If the answer was yes, what foods do you know how to cook? Preparation capacity Does it have a kitchen equipped with a stove? Yes / No |
| If the answer was yes, what foods do you know how to cook? Preparation capacity Does it have a kitchen equipped with a stove? Yes / No |
| Preparation capacity Does it have a kitchen equipped with a stove? Yes / No |
| Does it have a kitchen equipped with a stove? Yes / No |
| Dose it have a kitchen equipped with a refrigerator? |
| Does it have a kitchen equipped with a ferrigerator? |
| Does it have a kitchen equipped with an oven? Yes / No |
| Opportunity |
| Time to eat |
| How many minutes a day do you have for breakfast? |
| How many minutes a day do you have to eat? |
| How many minutes a day do you have for dinner? |
| How many minutes a day do you have to consume snacks? |
| Prepare food |
| How many minutes a day do you have to prepare your breakfast? |
| How many minutes a day do you have to prepare your food? |
| How many minutes a day do you have to prepare your dinner? |
| How many minutes a day do you have to prepare your snacks? |
| Access to food |
| Are there places selling fresh food (fruits, vegetables) near your home? Yes / No / I do not know |
| Are there non-perishable food outlets near your home (beans, oatmeal, rice, crackers, etc.? Yes / No / I do not know |
| Food storage |
| Do you have a refrigerator at home? Yes / No |
| Do you have containers to store food (tupers)? Yes / No |
| Motivation |
| You want to change your eating habits |
| Would you like to improve your eating habits? Yes / No / I do not know |
| Would you like to eat healthier? Yes / No / I do not know |
| Would you like to be a more physically active person? Yes / No / I do not know |
| Emotions involved in your food consumption |

| Do you eat more food or less food when you are sad, angry, or happy? | Please specify the emotion and the effect it has on your hunger and satiety |
|---|---|
| Habits you are willing to char | , , , , , |
| Please write down the eating habits that you would be willing to change, for example, eat more fruits and vegetables, eat less beef, etc. | |
| Reasons for sustainable food const | umption |
| Please write how important the following aspects are to you when you are going to consume food 1 is not very important and 5 is very important | |
| Animal welfare | |
| Produced without animals suffering | (Not very important) 1 2 3 4 5 (Very important) |
| Produced in an animal-friendly way | (Not very important) 1 2 3 4 5 (Very important) |
| It is produced respecting the rights of animals | (Not very important) 1 2 3 4 5 (Very important) |
| Produced with enough space for animals | (Not very important) 1 2 3 4 5 (Very important) |
| It is a free range or free range product | (Not very important) 1 2 3 4 5 (Very important) |
| Ethical concern | |
| Produced without exploitation | (Not very important) 1 2 3 4 5 (Very important) |
| Produced without child labor | (Not very important) 1 2 3 4 5 (Very important) |
| Traded fairly | (Not very important) 1 2 3 4 5 (Very important) |
| Environmental welfare | |
| Produced in an environmentally friendly way | (Not very important) 1 2 3 4 5 (Very important) |
| It is produced without disturbing the balance of nature | (Not very important) 1 2 3 4 5 (Very important) |
| Produced with minimal CO2 emissions | (Not very important) 1 2 3 4 5 (Very important) |
| It is packaged in an environmentally friendly way | (Not very important) 1 2 3 4 5 (Very important) |
| Local and seasonal | |
| It is a local/regional product | (Not very important) 1 2 3 4 5 (Very important) |
| It is a seasonal product | (Not very important) 1 2 3 4 5 (Very important) |
| It comes from nearby (short transport distance). | (Not very important) 1 2 3 4 5 (Very important) |

# Supplementary Material 5. Primers for bacteria identification in the qPCR analysis

| Bacteria | Name | Primer (5'-3') | Number of bases | Sequence | Notes | Reference |
|---|---|---|---|---|---|---|
| Firmicutes | 928F-Firm | Forward | 21 | 5'-TGAAACTCAAAGGAATTGACG-3' | $Y = C \text{ or } T \rightarrow C$ | |
| Firmicutes | 1040FirmR | Reverse | 17 | 5'-ACCATGCACCACCTGTC-3' | | _ |
| D | 798cfbF | Forward | 20 | 5'-CAAACAGGATTAGATACCCT-3' | $R = A \text{ or } G \rightarrow A$ | - (4.60) |
| Bacteroidetes | Cfb967R | Reverse | 19 | 5'-GGTAAGGTTCCTCGCGTAT-3' | | (4,68) |
| Universal | 926F | Forward | 20 | 5'-AAACTCAAAGGAATTGACGG-3' | $K = G \text{ or } T \rightarrow G$ | |
| Universal | 1062R | Reverse | 18 | 5'-CTCACAACACGAGCTGAC-3' | $R = A \text{ or } G \rightarrow A$ | |
| Lactobacillus | | Forward | 19 | 5'-AGCAGTAGGGAATCTTCCA-3' | | _ |
| Laciobacillus | | Reverse | 17 | 5'-CACCGCTACACATGGAG-3' | | <del>-</del> (70) |
| Difidah a atawiwa | | Forward | 18 | 5'-TCGCGTCCGGTGTGAAAG-3' | С | (70) |
| Бізіаодасіегіит | Bifidobacterium Reverse | | 17 | 5'-CCACATCCAGCATCCAC-3' | A | _ |
| Faecalibacterium | FPR-2F | Forward | 19 | 5'-GGAGGAAGAAGGTCTTCGG-3' | Amplicon 248 | <del>-</del> (73) |
| prausnitzii | Fprau645R | Reverse | 21 | 5'-AATTCCGCCTACCTCTGCACT-3' | | (73) |
| Akkermansia | | Forward | 20 | 5'-CAGCACGTGAAGGTGGGGAC-3' | | (74) |
| muciniphila | | Reverse | 20 | 5'-CCTTGCGGTTGGCTTCAGAT-3' | | - (74) |
| Duquotolla oonni | | Forward | 20 | 5'-CCGGACTCCTGCCCCTGCAA-3' | | (75) |
| Prevotella copri | | Reverse | 20 | 5'-GTTGCGCCAGGCACTGCGAT-3' | | <b>-</b> (75) |
| Bilophila | | Forward | 26 | 5'-CAACGTCCCCACCATCAAGTTCTCTG-3' | | (77) |
| wadsworthia | | Reverse | 26 | 5'-TGAATTCGCGGAAGGAGCGAGAGGTC-3' | | |
| Clostridium | | Forward | 19 | 5'-CGGTACCTGACTAAGAAGC-3' | 429 pb | _ |
| coccoides (Eubacterium rectale group and Lachnospiraceae family) | | Reverse | 19 | 5'-AGTTTCATTCTTGCGAACG-3' | 429 pb | (48) |
| Streptococcus | St1 | Forward | 22 | 5'-TTATTTGAAAGGGGCAATTGCT-3' | Posición: 195–216 | (90) |
| thermophilus | St2 | Reverse | 21 | 5'-GTGAACTTTCCACTCTCACAC-3' | Posición: 474–454 | <b>-</b> (80) |

Bases modified according to "Re: What are Y, M, W and D in primer design?", by A. Gund, Nadine, 2014. <a href="https://www.researchgate.net/post/What are Y M W and D in primer design/538c1577d11b8ba27a8b45df/citation/download">https://www.researchgate.net/post/What are Y M W and D in primer design/538c1577d11b8ba27a8b45df/citation/download</a>.

## Supplementary Material 6. Adherence questionnaire

This questionnaire will be updated based on the food plans to be designed, so the recommendations provided, and the consumption of the population will be contrasted, after the pilot test of this study. However, the format to be used and the questions developed so far are presented below.

Table SM6.1. Questionnaire of adherence to the sustainable-psycho-nutritional program

| Questionnaire of adherence to the sus | tainable | e-psvch | o-nutr | itiona | al pro | gram | | |
|---|---|---|---|---|---|---|---|---|
| Participant number: | | pojen | | - | vi pro | 9 | | |
| Date: | | | | | | | | |
| | Times per week | | | | | | | Times per day |
| Questions about food consumption | | 2 | 3 | 4 | 5 | 6 | 7 | |
| How many times a week do you eat foods that include corn? | | | | | | | | |
| How many times a week do you eat foods that include | | | | | | | | |
| amaranth? | | | | | | | | |
| How many times a week do you eat fruit? | | | | | | | | |
| How many times a week do you eat vegetables? | | | | | | | | |
| How many times a week do you eat foods that include beans? | | | | | | | | |
| How many times a week do you eat foods that include lentils? | | | | | | | | |
| How many times a week do you eat foods that include canola, | | | | | | | | |
| olive, or avocado oil? | | | | | | | | |
| How many times a week do you eat foods that include milk? | | | | | | | | |
| How many times a week do you eat foods that include cheese? | | | | | | | | |
| How many times a week do you eat foods that include yogurt? | | | | | | | | |
| How many times a week do you eat foods that include eggs? | | | | | | | | |
| How many times a week do you eat foods that include fish or | | | | | | | | |
| shellfish such as shrimp, octopus or crab? How many times a week do you eat foods that include | | | | | | | | |
| chicken? | | | | | | | | |
| How many times a week do you eat foods that include beef or | | | | | | | | |
| red meat such as pork, lamb, and goat? | | | | | | | | |
| How many times a week do you eat foods that include | | | | | | | | |
| processed meats like ham and sausage? | | | | | | | | |
| How many times a week do you consume soft drinks? | | | | | | | | |
| How many times a week do you eat packaged (ultra- | | | | | | | | |
| processed) foods? | | | | | | | | |
| Question about consumption reasons | | | | swers | | | | |
| Have you ever preferred to eat a particular food because of its | Yes | No | Explain your answer | | | | | |
| environmental impact? | | | pleas | se: | | | | |
| Have you ever preferred to eat a particular food because of its | Yes | No | Expl | loin | your | | swer | |
| impact on health and nutrition? | 1 68 | INO | pleas | | youi | an | SWCI | |
| impact on hearth and nutrition? | | | pica | | | | | |
| From 1 to 10, how much would you say you consumed the | Yes | No | | Explain your answer | | swer | | |
| meal plan that was provided to you? | | | pleas | se: | | | | |
| W 4 C 141-4 411 411 411 141 C 111 | 37 | NI- | T 1 | 1 | | | | |
| Was there any food that you did not like and therefore did not | Yes | No | Expl | | your | an | swer | |
| consume it? | | | pleas | sc. | | | | |

#### **Informed consent for study participants:**





Sustainable-psycho-nutritional intervention program and its effects on water and carbon footprint, metabolic biomarkers, and gut microbiota in Mexican population: study protocol of a m-Health randomized clinical trial

#### Brief Title:

stainable-psycho-nutritional intervention program and its effects on health outcomes and the environment

### Responsible institution:



Research Institute in Eating Behavior and Nutrition (Instituto de Investigaciones en Comportamiento Alimentario y Nutrición (IICAN), University Center of the South, University of Guadalajara. Address: Av. Enrique Arreola Silva 883, Col. Centro. Zip Code: 49000, Cd. Guzmán, Jalisco, México.

#### Collaborating institutions:



Institute of Nutrition and Food Technology "José Mataix Verdú", Biomedical Research Center, University of Granada, Avenida del Conocimiento S/N. Parque Tecnológico de la Salud. Armilla,18071 Granada, Spain



National Technological Institute of Mexico (Tecnológico Nacional de México, Campus Ciudad Guzmán) Address: Avenida Tecnológico 100, Col. Centro. Zip Code: 49000. Ciudad Guzmán, México.

Zapotlán el Grande, Jalisco. Date:



| By means of the present, I, I agree to |
|---|
| participate in the research project entitled: "Sustainable-psycho-nutritional intervention program and its |
| effects on water and carbon footprint, metabolic biomarkers, and gut microbiota in Mexican population: |
| study protocol of a m-Health randomized clinical trial". I am aware that the objective of this study is to design |
| a sustainable-psycho-nutritional intervention program and evaluate its effect on biological and environmental |
| indicators in the Mexican population. and that the information collected will be analyzed for non-profit research |
| purposes which will lead to publications in scientific journals. In addition, I am aware that at no time will I receive |

financial remuneration for my participation. I have been informed that my participation will consist of an evaluation of the following aspects. Anthropometric data: weight, height, waist and hip circumference. To do this I must take off my shoes and uncover my waist for less than 3 minutes. Biochemical data: blood sample and stool. For this, a specialist will take blood from my arm, so I will have to discover it and maintain a 12-hour overnight fast. Likewise, I will be given a sterile container to place a 3 cm<sup>3</sup> stool sample that I could be asked to preserve at the fridge if I a am not able to deliver it to the researcher as soon as I collected it. Clinical data: blood pressure measurement and superficial examination (e.g., face, neck, feet, hands), so I will uncover my left arm and allow the specialist to check my eyes, nails, hair, neck, and mouth, and, if necessary, the folds of my armpits. Dietary data: completion of dietary records and food frequency questionnaire. So, I will report the amounts of food I consume per day and on average per week, month, or year. I will be asked to write it down in paper, a mobile application, or a computer. Also, I may be asked to send photos of my food intake or uploaded into a mobile application. I am also aware that I will respond to a survey where I will provide sociodemographic and socioeconomic data, such as my educational level, my employment, a range of monthly income in Mexican pesos, among other data. In addition, I have been informed that I will have to use a mobile application that will help me improve my diet, both in relation to my nutrition and the environment. I know that the intervention in which I agree to participate will last 15 weeks, in which I will allow the extraction of blood and measurement of my weight, waist, and hip circumference on three occasions, as well as the visual physical examination and the taking of my blood pressure. I also know that I will deliver stool samples on a weekly basis, during the 15 weeks and that within the mobile application that I will use, I will be asked to record my food consumption on a daily basis, incorporating photographs and specifying the amounts of food consumed.

Additionally, I know that I may not be involved in the study but only evaluated. In addition, I know that the intervention, if it is part of it, will last 7 weeks, and additionally, there will be a 7-week follow-up period where I will be told whether or not I will be able to use the mobile application.

I know that the study will be carried out at the Centro Universitario del Sur, specifically at the Institute for Research in Eating Behavior and Nutrition (IICAN), as well as at the Laboratory of Biomedicine and Biotechnology for Health. In addition, it has been explained to me that my participation in this study is voluntary and I will not receive any financial compensation for it. However, I know that, if I wish, I will be able to obtain a

psycho-nutritional-sustainable diagnosis, and furthermore, with my participation I will benefit from obtaining nutritional counseling at the end of the intervention.

Finally, I confirm that I have been informed that the responsible researchers will maintain the confidentiality of my personal data based on the guidelines established by the Federal Law on Protection of Personal Data Held by Private Parties.

Therefore, I declare that:

- 1. I have read or had read to me the information provided.
- 2. I have had the opportunity to ask and all my doubts and questions have been satisfactorily clarified.
- 3. I voluntarily consent to participate in this research.
- 4. I understand that I have the right to withdraw at any time I choose without it affecting me in any way.
- 5. I have been informed that my refusal to participate will not cause me any problems.
- 6. I have been informed that the researchers undertake to answer any questions I may have during and after the data collection process.
- 7. I am aware that the main investigator will provide me with a diagnosis of my nutritional status and will provide me with nutritional guidance, if I wish.
- 8. I am aware that measurements will be taken on my waist and hips, so I will have to uncover my abdomen. In addition, I know that I will have to remove my shoes, socks and metallic accessories, including the belt, earrings, among other artifacts, when the main researcher of the study asked me to do so, before getting on the scale to be weighed and before being measured on the stadiometer.
- 9. I consent to a blood sample being taken and am aware that I will submit a stool sample on a weekly basis.
- 10. I agree to allow my blood pressure to be taken, visual examination of my neck, eyes, mouth, hair, nails and, if applicable, armpit folds. I also agree to fill in the questionnaires that the main researcher provides me, always answering as honestly as possible.
- 11. I agree to use a mobile application where I know that I will provide information, which will be confidential, but will help me improve my diet, both in relation to my nutrition and the environment. Likewise, and if I wish, I will be able to interact with other users within the mobile application and thus provide us with support.
  - 12. I accept that my data will be used in this and future studies, where my identity will always be protected.

If you have doubts or queries regarding participation in this study, you can contact the researcher responsible for this study, Mtra. Mariana Lares Michel, who is a doctoral student at the Institute for Research in Eating Behavior and Nutrition (IICAN). Her contact details are as follows: Av. Enrique Arreola Silva 883, Centro, C.P. 49000, Cd. Guzmán, Jalisco, Mexico, telephone: 3411017629. email: <a href="mariana.lmichel@alumnos.udg.mx">mariana.lmichel@alumnos.udg.mx</a> Also, you can contact Dr. Fatima Ezzahra Housni, who is the responsible researcher for this study at ClinicalTrials.gov. Her contact details are as follows: Av. Enrique Arreola Silva 883, Centro, C.P. 49000, Cd. Guzmán, Jalisco, Mexico, Tel.: (+52) 341 5752222 ext. 46142. email: <a href="fatima.housni@cusur.udg.mx">fatima.housni@cusur.udg.mx</a>

| Sincerely |
|--------------------------------------------|
| Place and date |
| Name and signature of the participant |
| Telephone: |
| Email: |
| Name and signature of the Witness 1. |
| Name and signature of the Witness 1: |
| Address and telephone: |
| Type of relationship with the participant: |
| Name and signature of the Witness 2. |
| Name and signature of the Witness 2: |
| Address and telephone: |
| Type of relationship with the participant: |

| I have explained to the participant the objective, justification and benefits that their participation implies. In turn, I have | • |
|---|---|
| and benefits that their participation implies. In turn, I have<br>that he has made me. Finally, I declare that I respect the go | * · |
| human beings. | underlines and regulations corresponding to research on |
| Name and signature of the investigator | Name and signature of the applicator |